CLINICAL TRIAL: NCT00122681
Title: A Phase III, Double-blind, Randomized, Controlled, Multi-center Study to Evaluate the Efficacy of GlaxoSmithKline Biologicals. HPV-16/18 VLP AS04 Vaccine Compared to Hepatitis A Vaccine as Control in Prevention of Persistent HPV-16 or HPV-18 Cervical Infection and Cervical Neoplasia, Administered Intramuscularly According to a 0, 1, 6 Month Schedule in Healthy Females 15-25 Years of Age.
Brief Title: Human Papilloma Virus (HPV) Vaccine Efficacy Trial Against Cervical Pre-cancer in Young Adults With GlaxoSmithKline (GSK) Biologicals HPV-16/18
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 580299/008
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Results first posted 2010-01-20 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2017-08

CONDITIONS: Infections, Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cervarix Group (Experimental): Subjects received 3 doses of Cervarix™ (GSK Biologicals' human papillomavirus [HPV] vaccine) at Months 0, 1 and 6.
  Interventions: Biological: Cervarix™
- Havrix Group (Active Comparator): Subjects received 3 doses of GSK Biologicals' hepatitis A vaccine [HAV] (Havrix™-based investigational formulation) at Months 0, 1 and 6.
  Interventions: Biological: Havrix™-based investigational formulation

INTERVENTIONS:
Biological: Cervarix™ — Intramuscular injection, 3 doses
  Other Names: GSK Biologicals HPV 16/18 VLP/AS04 vaccine
  Arms: Cervarix Group
Biological: Havrix™-based investigational formulation — Intramuscular injection, 3 doses
  Arms: Havrix Group

SUMMARY:
Human Papilloma virus (HPV) are viruses that cause a common infection of the skin and genitals in men and women. Several types of HPV infection are transmitted by sexual activity and, in women, can infect the cervix (part of the uterus or womb). This infection often goes away by itself, but if it does not go away (this is called persistent infection), it can lead in women over a long period of time to cancer of the cervix. If a woman is not infected by HPV, it is very unlikely that she will get cervical cancer. This study will evaluate the efficacy of GSK Biologicals HPV 16/18 VLP/AS04 vaccine to prevent infection associated cervical pre-cancer and vaccine with HPV 16 or 18 and the vaccine safety, over 48 months, in young adolescents and women of 15/25 years of age at study start. Approximately 18.000 study subjects will either receive the HPV vaccine or a control vaccine (hepatitis A vaccine) administered intramuscularly according to a 0-1-6 month schedule.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
NOTE: Some 178 centers participate in this study. Given that the recruitment is completed, the researchers have listed one center per country in this website. If required, further details of centers available on request.

ELIGIBILITY:
Inclusion Criteria:

* A woman whom the investigator believes that she and/or her parents/legally acceptable representative can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits).
* A woman between, and including, 15 and 25 years of age at the time of the first vaccination.
* Written informed consent must be obtained from the subject prior to enrollment (for subjects below the legal age of consent, written informed consent must be obtained from a parent or legal guardian of the subject and, in addition, the subject should sign and personally date a written informed assent).
* Subject must be free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Subject must have a negative urine pregnancy test.
* Subject must be of non-childbearing potential or, if of childbearing potential, she must be abstinent or must be using adequate contraceptive precautions for 30 days prior to the first vaccination and must agree to continue such precautions for two months after completion of the vaccination series.
* Has had no more than 6 lifetime sexual partners prior to enrollment. This criterion may not be applicable in subjects less than 18 years of age, according to local regulatory/ethical requirements.
* Subject must have intact cervix.

Exclusion Criteria:

* Pregnant or breastfeeding. Women must be at least 3 months post-pregnancy and not breastfeeding to enter the study.
* A woman planning to become pregnant or planning to discontinue contraceptive precautions during approximately the first nine months of the study (Months 0-8).
* Previous administration of components of the investigational vaccine.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after (i.e. days 0-29) each dose of vaccine. Administration of some routine vaccines up to 8 days before each dose of study vaccine is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Previous vaccination against human papillomavirus (HPV).
* History of vaccination against Hepatitis A or a known clinical history of Hepatitis A disease.
* History of having had colposcopy or has planned a colposcopy to evaluate an abnormal cervical cytology (Pap smear) test.
* Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccines.
* Hypersensitivity to latex.
* Known acute or chronic, clinically significant pulmonary, cardiovascular, neurologic, hepatic or renal functional abnormality, as determined by previous physical examination or laboratory tests.
* History of chronic condition(s) requiring treatment.
* Received immunoglobulins and/or blood product within 90 days preceding enrollment. Enrollment will be deferred until the subject is outside of specified window.
* Acute disease at the time of enrolment.
* Heavy bleeding (menstruation or other) or heavy vaginal discharge in which a pelvic exam cannot be performed. Enrollment will be deferred until condition is resolved according to investigator's medical judgement.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18729 (Actual)
Dates: Start 2004-05-06 (Actual); Primary Completion 2006-11-03 (Actual); Study Completion 2009-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (116):
- United States (42):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Louisville, Colorado
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, New Bern, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Webster, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, Wenatchee, Washington
- Australia (6):
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Carlton, Melbourne, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Perth, Western Australia
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Leuven
- Brazil (3):
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Campinas, São Paulo
- Canada (11):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Beauport, Quebec
  - GSK Investigational Site, Montreal, Quebec
- Finland (18):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Kerava
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kouvola
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Lappeenranta
  - GSK Investigational Site, Mikkeli
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Rauma
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vaasa
- Germany (13):
  - GSK Investigational Site, Karlsruhe, Baden-Wurttemberg
  - GSK Investigational Site, Ravensburg, Baden-Wurttemberg
  - GSK Investigational Site, Rheinstetten, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Dietzenbach, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Nordhausen, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Italy (2):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
- GSK Investigational Site, Cuenavaca, Morelos, Mexico
- Philippines (6):
  - GSK Investigational Site, Cavite
  - GSK Investigational Site, Laguna
  - GSK Investigational Site, Las Piñas
  - GSK Investigational Site, Los Banos, Laguna
  - GSK Investigational Site, Makati City
  - GSK Investigational Site, Manila
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Móstoles
- GSK Investigational Site, Taipei, Taiwan
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (4):
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Waterloo, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Lehtinen M, Lagheden C, Luostarinen T, Eriksson T, Apter D, Bly A, Gray P, Harjula K, Heikkila K, Hokkanen M, Karttunen H, Kuortti M, Nieminen P, Nummela M, Paavonen J, Palmroth J, Petaja T, Pukkala E, Soderlund-Strand A, Veivo U, Dillner J. Human papillomavirus vaccine efficacy against invasive, HPV-positive cancers: population-based follow-up of a cluster-randomised trial. BMJ Open. 2021 Dec 30;11(12):e050669. doi: 10.1136/bmjopen-2021-050669. PMID 35149535
- [Derived] Welby S, Rosillon D, Feng Y, Borys D. Progression from human papillomavirus (HPV) infection to cervical lesion or clearance in women (18-25 years): Natural history study in the control arm subjects of AS04-HPV-16/18 vaccine efficacy study in China between 2008 and 2016. Expert Rev Vaccines. 2022 Mar;21(3):407-413. doi: 10.1080/14760584.2022.2021077. Epub 2022 Jan 24. PMID 34939897
- [Derived] Adhikari I, Eriksson T, Luostarinen T, Apter D, Lehtinen M. Is the risk of cervical atypia associated with the interval between menarche and the start of sexual activity? A population-based cohort study. BMJ Open. 2019 Sep 11;9(9):e030091. doi: 10.1136/bmjopen-2019-030091. PMID 31511286
- [Derived] Castellsague X, Paavonen J, Jaisamrarn U, Wheeler CM, Skinner SR, Lehtinen M, Naud P, Chow SN, Del Rosario-Raymundo MR, Teixeira JC, Palmroth J, de Carvalho NS, Germar MJ, Peters K, Garland SM, Szarewski A, Poppe WA, Romanowski B, Schwarz TF, Tjalma WA, Bosch FX, Bozonnat MC, Struyf F, Dubin G, Rosillon D, Baril L; HPV PATRICIA Study Group. Risk of first cervical HPV infection and pre-cancerous lesions after onset of sexual activity: analysis of women in the control arm of the randomized, controlled PATRICIA trial. BMC Infect Dis. 2014 Oct 30;14:551. doi: 10.1186/s12879-014-0551-y. PMID 25927224
- [Derived] Apter D, Wheeler CM, Paavonen J, Castellsague X, Garland SM, Skinner SR, Naud P, Salmeron J, Chow SN, Kitchener HC, Teixeira JC, Jaisamrarn U, Limson G, Szarewski A, Romanowski B, Aoki FY, Schwarz TF, Poppe WA, Bosch FX, Mindel A, de Sutter P, Hardt K, Zahaf T, Descamps D, Struyf F, Lehtinen M, Dubin G; HPV PATRICIA Study Group. Efficacy of human papillomavirus 16 and 18 (HPV-16/18) AS04-adjuvanted vaccine against cervical infection and precancer in young women: final event-driven analysis of the randomized, double-blind PATRICIA trial. Clin Vaccine Immunol. 2015 Apr;22(4):361-73. doi: 10.1128/CVI.00591-14. Epub 2015 Feb 4. PMID 25651922
- [Derived] Struyf F, Colau B, Wheeler CM, Naud P, Garland S, Quint W, Chow SN, Salmeron J, Lehtinen M, Del Rosario-Raymundo MR, Paavonen J, Teixeira JC, Germar MJ, Peters K, Skinner SR, Limson G, Castellsague X, Poppe WA, Ramjattan B, Klein TD, Schwarz TF, Chatterjee A, Tjalma WA, Diaz-Mitoma F, Lewis DJ, Harper DM, Molijn A, van Doorn LJ, David MP, Dubin G; HPV PATRICIA Study Group. Post hoc analysis of the PATRICIA randomized trial of the efficacy of human papillomavirus type 16 (HPV-16)/HPV-18 AS04-adjuvanted vaccine against incident and persistent infection with nonvaccine oncogenic HPV types using an alternative multiplex type-specific PCR assay for HPV DNA. Clin Vaccine Immunol. 2015 Feb;22(2):235-44. doi: 10.1128/CVI.00457-14. Epub 2014 Dec 24. PMID 25540273
- [Derived] Castellsague X, Naud P, Chow SN, Wheeler CM, Germar MJ, Lehtinen M, Paavonen J, Jaisamrarn U, Garland SM, Salmeron J, Apter D, Kitchener H, Teixeira JC, Skinner SR, Limson G, Szarewski A, Romanowski B, Aoki FY, Schwarz TF, Poppe WA, Bosch FX, de Carvalho NS, Peters K, Tjalma WA, Safaeian M, Raillard A, Descamps D, Struyf F, Dubin G, Rosillon D, Baril L. Risk of newly detected infections and cervical abnormalities in women seropositive for naturally acquired human papillomavirus type 16/18 antibodies: analysis of the control arm of PATRICIA. J Infect Dis. 2014 Aug 15;210(4):517-34. doi: 10.1093/infdis/jiu139. Epub 2014 Mar 8. PMID 24610876
- [Derived] Jaisamrarn U, Castellsague X, Garland SM, Naud P, Palmroth J, Del Rosario-Raymundo MR, Wheeler CM, Salmeron J, Chow SN, Apter D, Teixeira JC, Skinner SR, Hedrick J, Szarewski A, Romanowski B, Aoki FY, Schwarz TF, Poppe WA, Bosch FX, de Carvalho NS, Germar MJ, Peters K, Paavonen J, Bozonnat MC, Descamps D, Struyf F, Dubin GO, Rosillon D, Baril L; HPV PATRICIA Study Group. Natural history of progression of HPV infection to cervical lesion or clearance: analysis of the control arm of the large, randomised PATRICIA study. PLoS One. 2013 Nov 19;8(11):e79260. doi: 10.1371/journal.pone.0079260. eCollection 2013. PMID 24260180
- [Derived] Valve P, Lehtinen-Jacks S, Eriksson T, Lehtinen M, Lindfors P, Saha MT, Rimpela A, Angle S. LINDA - a solution-focused low-intensity intervention aimed at improving health behaviors of young females: a cluster-randomized controlled trial. BMC Public Health. 2013 Nov 4;13:1044. doi: 10.1186/1471-2458-13-1044. PMID 24188719
- [Derived] Howell-Jones R, Soldan K, Wetten S, Mesher D, Williams T, Gill ON, Hughes G. Declining genital Warts in young women in england associated with HPV 16/18 vaccination: an ecological study. J Infect Dis. 2013 Nov 1;208(9):1397-403. doi: 10.1093/infdis/jit361. PMID 24092908
- [Derived] Szarewski A, Skinner SR, Garland SM, Romanowski B, Schwarz TF, Apter D, Chow SN, Paavonen J, Del Rosario-Raymundo MR, Teixeira JC, De Carvalho NS, Castro-Sanchez M, Castellsague X, Poppe WA, De Sutter P, Huh W, Chatterjee A, Tjalma WA, Ackerman RT, Martens M, Papp KA, Bajo-Arenas J, Harper DM, Torne A, David MP, Struyf F, Lehtinen M, Dubin G. Efficacy of the HPV-16/18 AS04-adjuvanted vaccine against low-risk HPV types (PATRICIA randomized trial): an unexpected observation. J Infect Dis. 2013 Nov 1;208(9):1391-6. doi: 10.1093/infdis/jit360. PMID 24092907
- [Derived] Roset Bahmanyar E, Paavonen J, Naud P, Salmeron J, Chow SN, Apter D, Kitchener H, Castellsague X, Teixeira JC, Skinner SR, Jaisamrarn U, Limson GA, Garland SM, Szarewski A, Romanowski B, Aoki F, Schwarz TF, Poppe WA, De Carvalho NS, Harper DM, Bosch FX, Raillard A, Descamps D, Struyf F, Lehtinen M, Dubin G; HPV PATRICIA Study Group. Prevalence and risk factors for cervical HPV infection and abnormalities in young adult women at enrolment in the multinational PATRICIA trial. Gynecol Oncol. 2012 Dec;127(3):440-50. doi: 10.1016/j.ygyno.2012.08.033. Epub 2012 Aug 30. PMID 22940493
- [Derived] Lehtinen M, Paavonen J, Wheeler CM, Jaisamrarn U, Garland SM, Castellsague X, Skinner SR, Apter D, Naud P, Salmeron J, Chow SN, Kitchener H, Teixeira JC, Hedrick J, Limson G, Szarewski A, Romanowski B, Aoki FY, Schwarz TF, Poppe WA, De Carvalho NS, Germar MJ, Peters K, Mindel A, De Sutter P, Bosch FX, David MP, Descamps D, Struyf F, Dubin G; HPV PATRICIA Study Group. Overall efficacy of HPV-16/18 AS04-adjuvanted vaccine against grade 3 or greater cervical intraepithelial neoplasia: 4-year end-of-study analysis of the randomised, double-blind PATRICIA trial. Lancet Oncol. 2012 Jan;13(1):89-99. doi: 10.1016/S1470-2045(11)70286-8. Epub 2011 Nov 8. PMID 22075171
- [Derived] Wheeler CM, Castellsague X, Garland SM, Szarewski A, Paavonen J, Naud P, Salmeron J, Chow SN, Apter D, Kitchener H, Teixeira JC, Skinner SR, Jaisamrarn U, Limson G, Romanowski B, Aoki FY, Schwarz TF, Poppe WA, Bosch FX, Harper DM, Huh W, Hardt K, Zahaf T, Descamps D, Struyf F, Dubin G, Lehtinen M; HPV PATRICIA Study Group. Cross-protective efficacy of HPV-16/18 AS04-adjuvanted vaccine against cervical infection and precancer caused by non-vaccine oncogenic HPV types: 4-year end-of-study analysis of the randomised, double-blind PATRICIA trial. Lancet Oncol. 2012 Jan;13(1):100-10. doi: 10.1016/S1470-2045(11)70287-X. Epub 2011 Nov 8. PMID 22075170
- [Derived] Szarewski A, Poppe WA, Skinner SR, Wheeler CM, Paavonen J, Naud P, Salmeron J, Chow SN, Apter D, Kitchener H, Castellsague X, Teixeira JC, Hedrick J, Jaisamrarn U, Limson G, Garland S, Romanowski B, Aoki FY, Schwarz TF, Bosch FX, Harper DM, Hardt K, Zahaf T, Descamps D, Struyf F, Lehtinen M, Dubin G; HPV PATRICIA Study Group. Efficacy of the human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine in women aged 15-25 years with and without serological evidence of previous exposure to HPV-16/18. Int J Cancer. 2012 Jul 1;131(1):106-16. doi: 10.1002/ijc.26362. Epub 2011 Oct 23. PMID 21858807
- [Derived] Wacholder S, Chen BE, Wilcox A, Macones G, Gonzalez P, Befano B, Hildesheim A, Rodriguez AC, Solomon D, Herrero R, Schiffman M; CVT group. Risk of miscarriage with bivalent vaccine against human papillomavirus (HPV) types 16 and 18: pooled analysis of two randomised controlled trials. BMJ. 2010 Mar 2;340:c712. doi: 10.1136/bmj.c712. PMID 20197322
- [Derived] Paavonen J, Naud P, Salmeron J, Wheeler CM, Chow SN, Apter D, Kitchener H, Castellsague X, Teixeira JC, Skinner SR, Hedrick J, Jaisamrarn U, Limson G, Garland S, Szarewski A, Romanowski B, Aoki FY, Schwarz TF, Poppe WA, Bosch FX, Jenkins D, Hardt K, Zahaf T, Descamps D, Struyf F, Lehtinen M, Dubin G; HPV PATRICIA Study Group. Efficacy of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine against cervical infection and precancer caused by oncogenic HPV types (PATRICIA): final analysis of a double-blind, randomised study in young women. Lancet. 2009 Jul 25;374(9686):301-14. doi: 10.1016/S0140-6736(09)61248-4. Epub 2009 Jul 6. PMID 19586656
- [Derived] Paavonen J, Jenkins D, Bosch FX, Naud P, Salmeron J, Wheeler CM, Chow SN, Apter DL, Kitchener HC, Castellsague X, de Carvalho NS, Skinner SR, Harper DM, Hedrick JA, Jaisamrarn U, Limson GA, Dionne M, Quint W, Spiessens B, Peeters P, Struyf F, Wieting SL, Lehtinen MO, Dubin G; HPV PATRICIA study group. Efficacy of a prophylactic adjuvanted bivalent L1 virus-like-particle vaccine against infection with human papillomavirus types 16 and 18 in young women: an interim analysis of a phase III double-blind, randomised controlled trial. Lancet. 2007 Jun 30;369(9580):2161-2170. doi: 10.1016/S0140-6736(07)60946-5. PMID 17602732
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 580299/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 580299/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 580299/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 580299/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 580299/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 580299/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 580299/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 18729 subjects enrolled in the study, 64 subjects were not vaccinated. Within the 18665 subjects vaccinated, 21 subjects from 1 center were excluded from all analyses because of potential data discrepancies identified at this center. As a result, a total of 18644 subjects are reported as started in the participant flow.
Period: Overall Study
Arm/Group | Havrix Group | Cervarix Group
Started | 9325 | 9319
Completed | 7811 | 7798
Not Completed | 1514 | 1521
Not completed — Adverse Event | 20 | 16
Not completed — Lost to Follow-up | 1080 | 1097
Not completed — Protocol Violation | 7 | 10
Not completed — Withdrawal by Subject | 257 | 251
Not completed — Personal reasons | 150 | 147

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Havrix Group | Cervarix Group | Total
Number analyzed (Participants) | 9325 | 9319 | 18644
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.0 (3.12) | 20.0 (3.10) | 20.0 (3.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9325 | 9319 | 18644
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)2+ Associated With HPV-16 and/or -18 Cervical Infection in Subjects HPV DNA Negative and Seronegative at Baseline or Overall (Any Serostatus at Baseline)
Description: CIN2+ was defined as CIN grades 2 and 3, endocervical adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Detection was done in:
  1. DNA- and sero-: subjects HPV deoxyribonucleic acid (DNA) negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative (sero-) for HPV-16 and/or HPV-18 by Enzyme-linked Immunosorbent Assay (ELISA) at baseline (Month 0).
  2. Overall: subjects DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
Time Frame: Up to the moment when 36 cases of CIN2+ lesions associated with HPV-16 or HPV-18 infection had been detected, including at least 15 cases of CIN2+ associated with HPV-18 infection. Mean follow-up was 34.9 months post-dose 3
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, which included all evaluable subjects who had received 3 doses of study vaccine, who had a normal or low-grade cytology (i.e. negative or Atypical Squamous Cells of Undetermined Significance (ASC-US) or Low-grade Squamous Intraepithelial Lesion (LSIL)) at Month 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7767 | 7814
Participants
  HPV-16/18, DNA- & sero- subjects: number analyzed (Participants) | 7312 | 7344
  HPV-16/18, DNA- & sero- subjects | 56 | 4
  HPV-16, DNA- & sero- subjects: number analyzed (Participants) | 6165 | 6303
  HPV-16, DNA- & sero- subjects | 46 | 2
  HPV-18, DNA- & sero- subjects: number analyzed (Participants) | 6746 | 6794
  HPV-18, DNA- & sero- subjects | 15 | 2
  HPV-16/18, overall | 65 | 6
  HPV-16, overall: number analyzed (Participants) | 7276 | 7372
  HPV-16, overall | 54 | 4
  HPV-18, overall: number analyzed (Participants) | 7583 | 7645
  HPV-18, overall | 16 | 2
Statistical Analysis 1: Comparison: Havrix Group vs Cervarix Group; Vaccine efficacy against CIN2+ associated with HPV-16 or HPV-18 (by PCR) in HPV DNA negative and seronegative subjects at baseline, using conditional exact method. The VE was defined as follows: VE = 1-Rate Ratio (RR), where RR = incidence rate in HPV Group (vaccine)/ incidence rate in HAV Group (control); Incidence rate = n/T(per 100); n= number of subjects reporting at least one event in each group and T(years) = sum of follow-up period (censored at the first occurrence of an event) expressed; Test type: Superiority or Other; 1-Rate Ratio = 92.9, 95% CI 2-sided [79.9 to 98.3]
Statistical Analysis 2: Comparison: Havrix Group vs Cervarix Group; Vaccine efficacy against CIN2+ associated with HPV-16 (by PCR) in HPV DNA negative and seronegative subjects at baseline, using conditional exact method. The VE was defined as follows: VE = 1-Rate Ratio (RR), where RR = incidence rate in HPV Group (vaccine)/ incidence rate in HAV Group (control); Incidence rate = n/T(per 100); n= number of subjects reporting at least one event in each group and T(years) = sum of follow-up period (censored at the first occurrence of an event) expressed; Test type: Superiority or Other; 1-Rate Ratio = 95.7, 95% CI 2-sided [82.9 to 99.6]
Statistical Analysis 3: Comparison: Havrix Group vs Cervarix Group; Vaccine efficacy against CIN2+ associated with HPV-18 (by PCR) in HPV DNA negative and seronegative subjects at baseline, using conditional exact method. The VE was defined as follows: VE = 1-Rate Ratio (RR), where RR = incidence rate in HPV Group (vaccine)/ incidence rate in HAV Group (control); Incidence rate = n/T(per 100); n= number of subjects reporting at least one event in each group and T(years) = sum of follow-up period (censored at the first occurrence of an event) expressed; Test type: Superiority or Other; 1-Rate Ratio = 86.7, 95% CI 2-sided [39.7 to 98.7]
Statistical Analysis 4: Comparison: Havrix Group vs Cervarix Group; Vaccine efficacy against CIN2+ for HPV-16 or HPV-18 (by PCR) in HPV DNA negative subjects at baseline, regardless of initial serostatus, using conditional exact method. The VE was defined as follows: VE = 1-Rate Ratio (RR), where RR = incidence rate in HPV Group (vaccine)/ incidence rate in HAV Group (control); Incidence rate = n/T(per 100); n= number of subjects reporting at least one event in each group and T(years) = sum of follow-up period (censored at the first occurrence of an event); Test type: Superiority or Other; 1-Rate Ratio = 90.8, 95% CI 2-sided [78.1 to 96.9]
Statistical Analysis 5: Comparison: Havrix Group vs Cervarix Group; Vaccine efficacy against CIN2+ for HPV-16 (by PCR) in HPV DNA negative subjects at baseline, regardless of initial serostatus, using conditional exact method. The VE was defined as follows: VE = 1-Rate Ratio (RR), where RR = incidence rate in HPV Group (vaccine)/ incidence rate in HAV Group (control); Incidence rate = n/T(per 100); n= number of subjects reporting at least one event in each group and T(years) = sum of follow-up period (censored at the first occurrence of an event); Test type: Superiority or Other; 1-Rate Ratio = 92.7, 95% CI 2-sided [79.3 to 98.2]
Statistical Analysis 6: Comparison: Havrix Group vs Cervarix Group; Vaccine efficacy against CIN2+ for HPV-18 (by PCR) in HPV DNA negative subjects at baseline, regardless of initial serostatus, using conditional exact method. The VE was defined as follows: VE = 1-Rate Ratio (RR), where RR = incidence rate in HPV Group (vaccine)/ incidence rate in HAV Group (control); Incidence rate = n/T(per 100); n= number of subjects reporting at least one event in each group and T(years) = sum of follow-up period (censored at the first occurrence of an event); Test type: Superiority or Other; 1-Rate Ratio = 87.6, 95% CI 2-sided [44.1 to 98.8]

2. Primary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)2+ Associated With HPV-16 and/or -18 Cervical Infection in Subjects HPV DNA Negative and Seronegative at Baseline or Overall (Any Serostatus at Baseline)
Description: CIN2+ was defined as CIN grades 2 and 3, endocervical adenocarcinoma in situ (AIS) and invasive cervical cancer.
  Detection was done in subjects:
  1. DNA- and sero-: HPV deoxyribonucleic acid (DNA) negative (DNA-) at Month 0 and Month 6 for the corresponding HPV-type and seronegative (sero-) for HPV-16 and/or HPV-18 by Enzyme-linked Immunosorbent Assay (ELISA) at baseline (Month 0)
  2. Overall: subjects HPV DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline.
Time Frame: at Month 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7760 | 7806
Participants
  HPV-16/18, DNA- & sero- subjects: number analyzed (Participants) | 7305 | 7338
  HPV-16/18, DNA- & sero- subjects | 97 | 5
  HPV-16, DNA- & sero- subjects: number analyzed (Participants) | 6160 | 6296
  HPV-16, DNA- & sero- subjects | 81 | 2
  HPV-18, DNA- & sero- subjects: number analyzed (Participants) | 6739 | 6789
  HPV-18, DNA- & sero- subjects | 23 | 3
  HPV-16/18, overall | 108 | 7
  HPV-16, overall: number analyzed (Participants) | 7267 | 7364
  HPV-16, overall | 91 | 4
  HPV-18, overall: number analyzed (Participants) | 7577 | 7638
  HPV-18, overall | 24 | 3
Statistical Analysis 1: Comparison: Havrix Group vs Cervarix Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; 1-Rate Ratio = 94.9, 95% CI 2-sided [87.7 to 98.4]
Statistical Analysis 2: Comparison: Havrix Group vs Cervarix Group; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; 1-Rate Ratio = 97.6, 95% CI 2-sided [91.0 to 99.7]
Statistical Analysis 3: Comparison: Havrix Group vs Cervarix Group; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; 1-Rate Ratio = 87.1, 95% CI 2-sided [57.2 to 97.5]
Statistical Analysis 4: Comparison: Havrix Group vs Cervarix Group; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; 1-Rate Ratio = 93.6, 95% CI 2-sided [86.3 to 97.5]
Statistical Analysis 5: Comparison: Havrix Group vs Cervarix Group; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; 1-Rate Ratio = 95.7, 95% CI 2-sided [88.5 to 98.9]
Statistical Analysis 6: Comparison: Havrix Group vs Cervarix Group; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; 1-Rate Ratio = 87.6, 95% CI 2-sided [59.2 to 97.6]

3. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 or HPV-18 Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN1+ was defined as histopathologically-confirmed lesions including cervical intraepithelial neoplasia of grade 1 (CIN1), grade 2 (CIN2), grade 3 (CIN3), AIS and invasive cervical cancer.
  Detection was done in subjects:
  1. DNA- and sero-: subjects HPV DNA- at Month 0 and Month 6 for the corresponding HPV-type and sero- for HPV-16 and/or HPV-18 by Enzyme-linked Immunosorbent Assay (ELISA) at baseline (Month 0)
  2. Overall: subjects HPV DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline
Time Frame: Up to the moment when 36 cases of CIN2+ lesions associated with HPV-16 or HPV-18 infection had been detected, including at least 15 cases of CIN2+ associated with HPV-18 infection. Mean follow-up was 34.9 months post dose 3
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, which included all evaluable subjects, who had received 3 doses of study vaccine and who had a normal or low-grade cytology (i.e. negative or ASC-US or LSIL) at Month 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7767 | 7814
Participants
  HPV-16/18, DNA- & sero-: number analyzed (Participants) | 7312 | 7344
  HPV-16/18, DNA- & sero- | 96 | 8
  HPV-16, DNA- & sero-: number analyzed (Participants) | 6165 | 6303
  HPV-16, DNA- & sero- | 70 | 5
  HPV-18, DNA- & sero-: number analyzed (Participants) | 6746 | 6794
  HPV-18, DNA- & sero- | 31 | 3
  HPV-16/18, overall | 111 | 12
  HPV-16, overall: number analyzed (Participants) | 7276 | 7372
  HPV-16, overall | 84 | 9
  HPV-18, overall: number analyzed (Participants) | 7583 | 7645
  HPV-18, overall | 32 | 3

4. Secondary Outcome: Number of Subjects Reporting Solicited Local and General Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Solicited general symptoms assessed include arthralgia, fatigue, fever (measured in degree celsius (°C) by axillary route), gastrointestinal symptoms, headache, myalgia, rash and urticaria.
  Data are presented across the 3 doses.
Time Frame: Within 7 days after any vaccination
Population: Analysis was performed on a safety subset of the Total vaccinated cohort, which included vaccinated subjects from certain sites. Data are presented for the total subset (total), then stratified subject HPV-16/18 DNA & serostatus at baseline: DNA positive (DNA+) or negative (DNA-), ELISA seropositive (sero+) or seronegative (sero-).
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 3081 | 3078
Participants
  Pain, total: number analyzed (Participants) | 3080 | 3078
  Pain, total | 2403 | 2787
  Pain, sero+ or DNA+: number analyzed (Participants) | 827 | 830
  Pain, sero+ or DNA+ | 622 | 743
  Pain, sero- & DNA-: number analyzed (Participants) | 2219 | 2211
  Pain, sero- & DNA- | 1758 | 2013
  Pain, DNA+: number analyzed (Participants) | 212 | 236
  Pain, DNA+ | 166 | 219
  Redness, total: number analyzed (Participants) | 3080 | 3078
  Redness, total | 851 | 1349
  Redness, sero+ or DNA+: number analyzed (Participants) | 827 | 830
  Redness, sero+ or DNA+ | 211 | 335
  Redness, sero- & DNA-: number analyzed (Participants) | 2219 | 2211
  Redness, sero- & DNA- | 630 | 1005
  Redness, DNA+: number analyzed (Participants) | 212 | 236
  Redness, DNA+ | 56 | 96
  Swelling, total: number analyzed (Participants) | 3080 | 3078
  Swelling, total | 609 | 1293
  Swelling, sero+ or DNA+: number analyzed (Participants) | 827 | 830
  Swelling, sero+ or DNA+ | 145 | 325
  Swelling, sero- & DNA-: number analyzed (Participants) | 2219 | 2211
  Swelling, sero- & DNA- | 454 | 959
  Swelling, DNA+: number analyzed (Participants) | 212 | 236
  Swelling, DNA+ | 27 | 93
  Arthralgia, total | 551 | 633
  Arthralgia, sero+ or DNA+: number analyzed (Participants) | 828 | 830
  Arthralgia, sero+ or DNA+ | 160 | 149
  Arthralgia, sero- & DNA-: number analyzed (Participants) | 2219 | 2211
  Arthralgia, sero- & DNA- | 384 | 480
  Arthralgia, DNA+: number analyzed (Participants) | 212 | 236
  Arthralgia, DNA+ | 39 | 58
  Fatigue, total | 1652 | 1771
  Fatigue, sero+ or DNA+: number analyzed (Participants) | 828 | 830
  Fatigue, sero+ or DNA+ | 415 | 443
  Fatigue, sero- & DNA-: number analyzed (Participants) | 2219 | 2211
  Fatigue, sero- & DNA- | 1215 | 1311
  Fatigue, DNA+: number analyzed (Participants) | 212 | 236
  Fatigue, DNA+ | 116 | 123
  Fever ≥ 37.5°C, total | 342 | 385
  Fever ≥ 37.5°C, sero+ or DNA+: number analyzed (Participants) | 828 | 830
  Fever ≥ 37.5°C, sero+ or DNA+ | 103 | 126
  Fever ≥ 37.5°C, sero- & DNA-: number analyzed (Participants) | 2219 | 2211
  Fever ≥ 37.5°C, sero- & DNA- | 236 | 254
  Fever ≥ 37.5°C, DNA+: number analyzed (Participants) | 212 | 236
  Fever ≥ 37.5°C, DNA+ | 23 | 37
  Gastro-intestinal symptoms, total | 847 | 856
  Gastro-intestinal,sero+ or DNA+: number analyzed (Participants) | 828 | 830
  Gastro-intestinal,sero+ or DNA+ | 241 | 248
  Gastro-intestinal,sero- & DNA-: number analyzed (Participants) | 2219 | 2211
  Gastro-intestinal,sero- & DNA- | 595 | 601
  Gastro-intestinal symptoms, DNA+: number analyzed (Participants) | 212 | 236
  Gastro-intestinal symptoms, DNA+ | 64 | 72
  Headache, total | 1583 | 1668
  Headache, sero+ or DNA+: number analyzed (Participants) | 828 | 830
  Headache, sero+ or DNA+ | 423 | 425
  Headache, sero- & DNA-: number analyzed (Participants) | 2219 | 2211
  Headache, sero- & DNA- | 1141 | 1223
  Headache, DNA+: number analyzed (Participants) | 212 | 236
  Headache, DNA+ | 112 | 125
  Myalgia, total | 1381 | 1607
  Myalgia, sero+ or DNA+: number analyzed (Participants) | 828 | 830
  Myalgia, sero+ or DNA+ | 347 | 392
  Myalgia, sero- & DNA-: number analyzed (Participants) | 2219 | 2211
  Myalgia, sero- & DNA- | 1019 | 1200
  Myalgia, DNA+: number analyzed (Participants) | 212 | 236
  Myalgia, DNA+ | 85 | 119
  Rash, total | 258 | 314
  Rash, sero+ or DNA+: number analyzed (Participants) | 828 | 830
  Rash, sero+ or DNA+ | 72 | 91
  Rash, sero- & DNA-: number analyzed (Participants) | 2219 | 2211
  Rash, sero- & DNA- | 182 | 221
  Rash, DNA+: number analyzed (Participants) | 212 | 236
  Rash, DNA+ | 19 | 29
  Urticaria, total | 244 | 300
  Urticaria, sero+ or DNA+: number analyzed (Participants) | 828 | 830
  Urticaria, sero+ or DNA+ | 73 | 90
  Urticaria, sero- & DNA-: number analyzed (Participants) | 2219 | 2211
  Urticaria, sero- & DNA- | 169 | 206
  Urticaria, DNA+: number analyzed (Participants) | 212 | 236
  Urticaria, DNA+ | 14 | 25

5. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events
Description: Unsolicited adverse event (AE) covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 30 days after any vaccination
Population: Analysis was performed on the Safety Subset of the Total Vaccinated Cohort and stratified according to initial (Month 0) HPV-16/18 DNA Status and According to HPV-16 or -18 Serostatus.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 3187 | 3184
Participants
  total | 1466 | 1448
  sero+ DNA+: number analyzed (Participants) | 858 | 854
  sero+ DNA+ | 400 | 386
  sero- DNA-: number analyzed (Participants) | 2289 | 2290
  sero- DNA- | 1048 | 1049
  DNA+: number analyzed (Participants) | 222 | 243
  DNA+ | 111 | 122

6. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the entire study period (Month 0 to Month 48)
Population: Analysis was performed on the Total Vaccinated Cohort. The data are presented stratified by initial (Month 0) HPV-16/18 DNA status and according to HPV-16 or 18 serostatus (by ELISA).
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 9325 | 9319
Participants
  Total | 829 | 835
  Sero + and DNA +: number analyzed (Participants) | 2419 | 2409
  Sero + and DNA + | 239 | 251
  Sero- and DNA-: number analyzed (Participants) | 6789 | 6804
  Sero- and DNA- | 587 | 576
  DNA+: number analyzed (Participants) | 649 | 690
  DNA+ | 69 | 82

7. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Disease (NOCDs)
Description: NOCDs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: Throughout the entire study (Month 0 to 48)
Population: Analysis was performed on the Total Vaccinated Cohort and stratified according to initial (Month 0) HPV-16/18 DNA Status and According to HPV-16 or -18 Serostatus.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 9325 | 9319
Participants
  Total | 307 | 285
  sero+ and DNA+: number analyzed (Participants) | 2419 | 2409
  sero+ and DNA+ | 79 | 79
  sero- and DNA-: number analyzed (Participants) | 6789 | 6804
  sero- and DNA- | 225 | 201
  DNA+: number analyzed (Participants) | 649 | 690
  DNA+ | 21 | 24

8. Secondary Outcome: Number of Subjects Reporting Medically Significant Conditions
Description: Medically significant conditions include adverse events (AEs) prompting emergency room or physician visits that are not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that are not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: Throughout entire study period (Month 0 to Month 48)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 9325 | 9319
Participants
  Total | 3378 | 3298
  sero+ DNA+: number analyzed (Participants) | 2419 | 2409
  sero+ DNA+ | 957 | 958
  sero- DNA-: number analyzed (Participants) | 6789 | 6804
  sero- DNA- | 2378 | 2303
  DNA+: number analyzed (Participants) | 649 | 690
  DNA+ | 285 | 296

9. Secondary Outcome: Number of Subjects With Outcome of Pregnancies, Overall and Stratified by Initial (Month 0) HPV-16/18 DNA Status and According to HPV-16 or -18 Serostatus
Description: Pregnancy outcomes are normal infant, premature infant, abnormal infant, elective termination, therapeutic abortion, ectopic pregnancy, spontaneous abortion, still birth, lost to follow-up, no pregnancy/molar pregnancy, pregnancy ongoing.
Time Frame: Throughout the entire study period (Month 0 to Month 48)
Population: as for outcome 7
Measure: Number; unit: subjects
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 2257 | 2257
subjects
  total, normal infant | 1671 | 1642
  total, premature birth | 66 | 77
  total, abnormal infant | 22 | 26
  total, elective termination | 228 | 212
  total, therapeutic abortion | 1 | 2
  total, ectopic pregnancy | 9 | 20
  total, spontaneous abortion | 195 | 205
  total, still birth | 11 | 16
  total, lost to follow-up | 42 | 41
  total, no pregnancy, molar pregnancy | 1 | 4
  total, pregnancy ongoing | 11 | 12
  sero- DNA- (n=1553, 1540), normal infant: number analyzed (Participants) | 1553 | 1540
  sero- DNA- (n=1553, 1540), normal infant | 1164 | 1159
  sero- DNA-, premature birth | 42 | 37
  sero- DNA-, abnormal infant | 15 | 18
  sero- DNA-, elective termination | 162 | 138
  sero- DNA-, therapeutic abortion | 0 | 1
  sero- DNA-, ectopic pregnancy | 7 | 13
  sero- DNA-, spontaneous abortion | 125 | 134
  sero- DNA -, still birth | 8 | 10
  sero- DNA-, lost to follow-up | 21 | 21
  sero- DNA-, no pregnancy, molar pregnancy | 1 | 3
  sero- DNA-, pregnancy ongoing | 8 | 6
  sero+ DNA+, normal infant | 486 | 464
  sero+ DNA+, premature birth | 24 | 39
  sero+ DNA+, abnormal infant | 6 | 8
  sero+ DNA+, elective termination | 62 | 67
  sero+ DNA+, therapeutic abortion | 1 | 1
  sero+ DNA+, ectopic pregnancy | 2 | 7
  sero+ DNA+, spontaneous abortion | 68 | 67
  sero+ DNA+, still birth | 3 | 6
  sero+ DNA+, lost to follow-up | 21 | 19
  sero+ DNA+, no pregnancy, molar pregnancy | 0 | 1
  sero+ DNA+, pregnancy ongoing | 3 | 6
  DNA+(n=162, 199), normal infant | 110 | 131
  DNA+, premature infant | 5 | 19
  DNA+, abnormal infant | 0 | 0
  DNA+, elective termination | 21 | 18
  DNA+, therapeutic abortion | 0 | 1
  DNA+, ectopic pregnancy | 0 | 2
  DNA+, spontaneous abortion | 18 | 21
  DNA+, still birth | 0 | 1
  DNA+, lost to follow-up | 7 | 5
  DNA+, no pregnancy, molar pregnancy | 0 | 0
  DNA+, pregnancy ongoing | 1 | 1

10. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With HPV-16 or HPV-18
Description: Persistent cervical HPV infection (6-month definition) was defined as the detection of the same HPV type by polymerase chain reaction (PCR) in cervical samples at 2 consecutive evaluations over approximately a 6-month interval.
  Detection was done in subjects:
  1. DNA- and sero-: subjects HPV DNA- at Month 0 and Month 6 for the corresponding HPV-type and sero- for HPV-16 and/or HPV-18 by Enzyme-linked Immunosorbent Assay (ELISA) at baseline (Month 0)
  2. Overall: subjects HPV DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline
Time Frame: as for outcome 3
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, which included all evaluable subjects, who had received 3 doses of study vaccine and who had a normal or low-grade cytology (i.e. negative or ASC-US or LSIL) at Month 0. All subjects had at least 5 months of follow-up after Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7556 | 7619
Participants
  HPV-16/18, DNA- & sero-: number analyzed (Participants) | 7122 | 7177
  HPV-16/18, DNA- & sero- | 488 | 29
  HPV-16, DNA- & sero-: number analyzed (Participants) | 6018 | 6163
  HPV-16, DNA- & sero- | 337 | 22
  HPV-18, DNA- & sero-: number analyzed (Participants) | 6567 | 6642
  HPV-18, DNA- & sero- | 184 | 7
  HPV-16/18, overall | 540 | 37
  HPV-16, overall: number analyzed (Participants) | 7085 | 7196
  HPV-16, overall | 380 | 29
  HPV-18, overall: number analyzed (Participants) | 7377 | 7457
  HPV-18, overall | 195 | 8

11. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With HPV-16 or HPV-18
Description: as for outcome 10
Time Frame: at Month 48
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, which included all evaluable subjects, who had received 3 doses of study vaccine, who had a normal or low-grade cytology (i.e. negative or ASC-US or LSIL) at Month 0. All subjects had at least 5 months of follow-up after Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7572 | 7626
Participants
  HPV-16/18, DNA- & sero-: number analyzed (Participants) | 7137 | 7182
  HPV-16/18, DNA- & sero- | 588 | 35
  HPV-16, DNA- & sero-: number analyzed (Participants) | 6029 | 6165
  HPV-16, DNA- & sero- | 418 | 24
  HPV-18, DNA- & sero-: number analyzed (Participants) | 6581 | 6649
  HPV-18, DNA- & sero- | 212 | 11
  HPV-16/18, overall | 654 | 45
  HPV-16, overall: number analyzed (Participants) | 7099 | 7202
  HPV-16, overall | 473 | 31
  HPV-18, overall: number analyzed (Participants) | 7394 | 7465
  HPV-18, overall | 227 | 14

12. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Oncogenic HPV Types
Description: Oncogenic types included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Detection was done in subjects who were HPV DNA negative at baseline regardless of initial serostatus.
  HRW-HPV= All high-risk (oncogenic) HPV types excluding HPV-16 and HPV-18 HR-HPV= High-risk (oncogenic) HPV types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68
Time Frame: as for outcome 3
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7640 | 7665
Participants
  HPV-16: number analyzed (Participants) | 7085 | 7196
  HPV-16 | 380 | 29
  HPV-18: number analyzed (Participants) | 7377 | 7457
  HPV-18 | 195 | 8
  HPV-31: number analyzed (Participants) | 7398 | 7394
  HPV-31 | 199 | 45
  HPV-33: number analyzed (Participants) | 7496 | 7527
  HPV-33 | 100 | 55
  HPV-35: number analyzed (Participants) | 7553 | 7572
  HPV-35 | 43 | 55
  HPV- 39: number analyzed (Participants) | 7411 | 7423
  HPV- 39 | 149 | 147
  HPV-45: number analyzed (Participants) | 7540 | 7587
  HPV-45 | 79 | 19
  HPV-51: number analyzed (Participants) | 7152 | 7188
  HPV-51 | 354 | 304
  HPV-52: number analyzed (Participants) | 7221 | 7280
  HPV-52 | 315 | 293
  HPV-56: number analyzed (Participants) | 7435 | 7460
  HPV-56 | 174 | 182
  HPV-58: number analyzed (Participants) | 7494 | 7512
  HPV-58 | 101 | 111
  HPV-59: number analyzed (Participants) | 7514 | 7528
  HPV-59 | 59 | 56
  HPV-66: number analyzed (Participants) | 7358 | 7405
  HPV-66 | 178 | 168
  HPV-68: number analyzed (Participants) | 7409 | 7441
  HPV-68 | 134 | 138
  HRW-HPV | 1351 | 1207
  HR-HPV | 1607 | 1233

13. Secondary Outcome: Number of Subjects With Persistent Infection (6-month Definition) With Oncogenic HPV Types
Description: Oncogenic types included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Detection was done in subjects who were HPV DNA negative at baseline regardless of initial serostatus.
  HRW-HPV = All high-risk (oncogenic) HPV types excluding HPV-16 and HPV-18 HR-HPV = High-risk (oncogenic) HPV types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68
Time Frame: at Month 48
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7656 | 7672
Participants
  HPV-16: number analyzed (Participants) | 7099 | 7202
  HPV-16 | 473 | 31
  HPV-18: number analyzed (Participants) | 7394 | 7465
  HPV-18 | 227 | 14
  HPV-31: number analyzed (Participants) | 7414 | 7400
  HPV-31 | 247 | 58
  HPV-33: number analyzed (Participants) | 7513 | 7534
  HPV-33 | 117 | 65
  HPV-35: number analyzed (Participants) | 7569 | 7579
  HPV-35 | 56 | 67
  HPV-39: number analyzed (Participants) | 7428 | 7429
  HPV-39 | 184 | 175
  HPV-45: number analyzed (Participants) | 7556 | 7594
  HPV-45 | 90 | 24
  HPV-51: number analyzed (Participants) | 7165 | 7190
  HPV-51 | 416 | 349
  HPV-52: number analyzed (Participants) | 7237 | 7289
  HPV-52 | 374 | 346
  HPV-56: number analyzed (Participants) | 7451 | 7467
  HPV-56 | 215 | 226
  HPV-58: number analyzed (Participants) | 7511 | 7518
  HPV-58 | 122 | 144
  HPV-59: number analyzed (Participants) | 7530 | 7536
  HPV-59 | 68 | 73
  HPV-66: number analyzed (Participants) | 7375 | 7412
  HPV-66 | 215 | 211
  HPV-68: number analyzed (Participants) | 7424 | 7450
  HPV-68 | 169 | 165
  HRW-HPV | 1556 | 1399
  HR-HPV | 1837 | 1424

14. Secondary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With HPV-16 or HPV-18 Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 3
Time Frame: at Month 48
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, which included all evaluable subjects who had a normal or low-grade cytology (i.e. negative or ASC-US or LSIL) at Month 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7760 | 7806
Participants
  HPV-16/18, DNA- & sero-: number analyzed (Participants) | 7305 | 7338
  HPV-16/18, DNA- & sero- | 165 | 12
  HPV-16, DNA- & sero-: number analyzed (Participants) | 6160 | 6296
  HPV-16, DNA- & sero- | 124 | 6
  HPV-18, DNA- & sero-: number analyzed (Participants) | 6739 | 6789
  HPV-18, DNA- & sero- | 52 | 6
  HPV-16/18, overall | 182 | 16
  HPV-16, overall: number analyzed (Participants) | 7267 | 7364
  HPV-16, overall | 140 | 10
  HPV-18, overall: number analyzed (Participants) | 7577 | 7638
  HPV-18, overall | 53 | 6

15. Secondary Outcome: Number of Subjects Reporting Persistent Infection (12-month Definition) With HPV-16 or HPV-18
Description: Persistent cervical HPV infection (12-month definition) was defined as the detection of the same HPV type (by PCR) over a 12-month interval (evaluations were planned at approximately 6-month intervals).
  Detection was done in subjects:
  1. DNA- and sero-: subjects HPV DNA- at Month 0 and Month 6 for the corresponding HPV-type and sero- for HPV-16 and/or HPV-18 by Enzyme-linked Immunosorbent Assay (ELISA) at baseline (Month 0)
  2. Overall: subjects HPV DNA- at Month 0 and Month 6 for the corresponding HPV-type and regardless of initial serostatus at baseline
Time Frame: as for outcome 3
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy, which included all evaluable subjects, who had received 3 doses of study vaccine and who had a normal or low-grade cytology (i.e. negative or ASC-US or LSIL) at Month 0. All subjects had at least 10 months of follow-up after Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7404 | 7466
Participants
  HPV-16/18, DNA- & sero-: number analyzed (Participants) | 6984 | 7035
  HPV-16/18, DNA- & sero- | 227 | 20
  HPV-16, DNA- & sero-: number analyzed (Participants) | 5903 | 6052
  HPV-16, DNA- & sero- | 171 | 17
  HPV-18, DNA- & sero-: number analyzed (Participants) | 6440 | 6508
  HPV-18, DNA- & sero- | 66 | 3
  HPV-16/18, overall | 252 | 21
  HPV-16, overall: number analyzed (Participants) | 6941 | 7057
  HPV-16, overall | 192 | 18
  HPV-18, overall: number analyzed (Participants) | 7231 | 7307
  HPV-18, overall | 70 | 3

16. Secondary Outcome: Number of Subjects Reporting Persistent Infection (12-month Definition) With HPV-16 or HPV-18
Description: as for outcome 15
Time Frame: at Month 48
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7461 | 7517
Participants
  HPV-16/18, DNA- & sero-: number analyzed (Participants) | 7038 | 7082
  HPV-16/18, DNA- & sero- | 354 | 26
  HPV-16, DNA- & sero-: number analyzed (Participants) | 5949 | 6089
  HPV-16, DNA- & sero- | 269 | 19
  HPV-18, DNA- & sero-: number analyzed (Participants) | 6490 | 6552
  HPV-18, DNA- & sero- | 98 | 7
  HPV-16/18, overall | 388 | 28
  HPV-16, overall: number analyzed (Participants) | 6996 | 7103
  HPV-16, overall | 300 | 20
  HPV-18, overall: number analyzed (Participants) | 7288 | 7356
  HPV-18, overall | 103 | 8

17. Secondary Outcome: Number of Subjects With Histopathologically Confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With Oncogenic HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: Oncogenic HPV types assessed included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Detection was done in subjects who were HPV DNA negative at baseline regardless of initial serostatus.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7764 | 7782
Participants
  HPV-16: number analyzed (Participants) | 7276 | 7372
  HPV-16 | 84 | 9
  HPV-18: number analyzed (Participants) | 7583 | 7645
  HPV-18 | 32 | 3
  HPV-31: number analyzed (Participants) | 7599 | 7583
  HPV-31 | 49 | 6
  HPV-33: number analyzed (Participants) | 7706 | 7720
  HPV-33 | 34 | 21
  HPV-35: number analyzed (Participants) | 7764 | 7768
  HPV-35 | 13 | 4
  HPV-39: number analyzed (Participants) | 7614 | 7609
  HPV-39 | 29 | 18
  HPV-45: number analyzed (Participants) | 7745 | 7782
  HPV-45 | 12 | 1
  HPV-51: number analyzed (Participants) | 7352 | 7363
  HPV-51 | 57 | 42
  HPV-52: number analyzed (Participants) | 7414 | 7461
  HPV-52 | 44 | 29
  HPV-56: number analyzed (Participants) | 7638 | 7646
  HPV-56 | 26 | 23
  HPV-58: number analyzed (Participants) | 7702 | 7709
  HPV-58 | 34 | 11
  HPV-59: number analyzed (Participants) | 7723 | 7720
  HPV-59 | 12 | 8
  HPV-66: number analyzed (Participants) | 7564 | 7592
  HPV-66 | 24 | 15
  HPV-68: number analyzed (Participants) | 7614 | 7633
  HPV-68 | 22 | 11

18. Secondary Outcome: Number of Subjects With Histopathologically Confirmed Cervical Intraepithelial Neoplasia (CIN)1+ Associated With Oncogenic HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 17
Time Frame: at Month 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7757 | 7774
Participants
  HPV-16: number analyzed (Participants) | 7267 | 7364
  HPV-16 | 140 | 10
  HPV-18: number analyzed (Participants) | 7577 | 7638
  HPV-18 | 53 | 6
  HPV-31: number analyzed (Participants) | 7592 | 7575
  HPV-31 | 79 | 11
  HPV-33: number analyzed (Participants) | 7700 | 7712
  HPV-33 | 66 | 23
  HPV-35: number analyzed (Participants) | 7757 | 7760
  HPV-35 | 18 | 7
  HPV-39: number analyzed (Participants) | 7608 | 7602
  HPV-39 | 48 | 26
  HPV-45: number analyzed (Participants) | 7738 | 7774
  HPV-45 | 25 | 3
  HPV-51: number analyzed (Participants) | 7341 | 7356
  HPV-51 | 96 | 61
  HPV-52: number analyzed (Participants) | 7409 | 7455
  HPV-52 | 81 | 51
  HPV-56: number analyzed (Participants) | 7631 | 7638
  HPV-56 | 45 | 36
  HPV-58: number analyzed (Participants) | 7696 | 7701
  HPV-58 | 42 | 25
  HPV-59: number analyzed (Participants) | 7716 | 7713
  HPV-59 | 20 | 13
  HPV-66: number analyzed (Participants) | 7559 | 7583
  HPV-66 | 44 | 30
  HPV-68: number analyzed (Participants) | 7606 | 7626
  HPV-68 | 43 | 28

19. Secondary Outcome: Number of Subjects With Histopathologically Confirmed Cervical Intraepithelial Neoplasia (CIN)2+ Associated With Oncogenic HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: CIN2+ was defined as histopathologically-confirmed lesions including cervical intraepithelial neoplasia of grade 2 (CIN2), grade 3 (CIN3), AIS and invasive cervical cancer.
  Oncogenic types detected included HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
  Detection was done in subjects who were HPV DNA negative at baseline, regardless of initial serostatus.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7764 | 7782
Participants
  HPV-16: number analyzed (Participants) | 7276 | 7372
  HPV-16 | 54 | 4
  HPV-18: number analyzed (Participants) | 7583 | 7645
  HPV-18 | 16 | 2
  HPV-31: number analyzed (Participants) | 7599 | 7583
  HPV-31 | 25 | 2
  HPV-33: number analyzed (Participants) | 7706 | 7720
  HPV-33 | 25 | 12
  HPV-35: number analyzed (Participants) | 7764 | 7768
  HPV-35 | 6 | 1
  HPV-39: number analyzed (Participants) | 7614 | 7609
  HPV-39 | 10 | 3
  HPV-45: number analyzed (Participants) | 7745 | 7782
  HPV-45 | 4 | 0
  HPV-51: number analyzed (Participants) | 7352 | 7363
  HPV-51 | 27 | 10
  HPV-52: number analyzed (Participants) | 7414 | 7461
  HPV-52 | 14 | 12
  HPV-56: number analyzed (Participants) | 7638 | 7646
  HPV-56 | 10 | 4
  HPV-58: number analyzed (Participants) | 7702 | 7709
  HPV-58 | 17 | 6
  HPV-59: number analyzed (Participants) | 7723 | 7720
  HPV-59 | 4 | 1
  HPV-66: number analyzed (Participants) | 7564 | 7592
  HPV-66 | 10 | 4
  HPV-68: number analyzed (Participants) | 7614 | 7633
  HPV-68 | 11 | 5

20. Secondary Outcome: Number of Subjects With Histopathologically Confirmed Cervical Intraepithelial Neoplasia (CIN)2+ Associated With Oncogenic HPV Types Detected Within the Lesional Component of the Cervical Tissue Specimen
Description: as for outcome 19
Time Frame: at Month 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 7757 | 7774
Participants
  HPV-16: number analyzed (Participants) | 7267 | 7364
  HPV-16 | 91 | 4
  HPV-18: number analyzed (Participants) | 7577 | 7638
  HPV-18 | 24 | 3
  HPV-31: number analyzed (Participants) | 7592 | 7575
  HPV-31 | 40 | 5
  HPV-33: number analyzed (Participants) | 7700 | 7712
  HPV-33 | 41 | 13
  HPV-35: number analyzed (Participants) | 7757 | 7760
  HPV-35 | 8 | 3
  HPV-39: number analyzed (Participants) | 7608 | 7602
  HPV-39 | 16 | 4
  HPV-45: number analyzed (Participants) | 7738 | 7774
  HPV-45 | 11 | 2
  HPV-51: number analyzed (Participants) | 7341 | 7356
  HPV-51 | 46 | 21
  HPV-52: number analyzed (Participants) | 7409 | 7455
  HPV-52 | 33 | 24
  HPV-56: number analyzed (Participants) | 7631 | 7638
  HPV-56 | 13 | 7
  HPV-58: number analyzed (Participants) | 7696 | 7701
  HPV-58 | 21 | 15
  HPV-59: number analyzed (Participants) | 7716 | 7713
  HPV-59 | 5 | 1
  HPV-66: number analyzed (Participants) | 7559 | 7583
  HPV-66 | 16 | 7
  HPV-68: number analyzed (Participants) | 7606 | 7626
  HPV-68 | 15 | 11

21. Secondary Outcome: Number of Seropositive Subjects for Anti-HPV-16 and Anti-HPV-18 Antibody Titers by ELISA in the Immunogenicity Subset, According to Initial (Month 0) HPV-16 or HPV-18 Serostatus
Description: Cut-off values assessed for seropositivity include 8 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
  Results are presented for the total group and stratified according to initial (Month 0) HPV-16 or HPV-18 serostatus by ELISA - seronegative (sero-) or seropositive (sero+)
Time Frame: At Months 6, 7, 12, 24, 36 & 48
Population: The analyses were performed on the ATP cohort for immunogenicity on evaluable subjects for whom immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 898 | 1036
Participants
  HPV-16, sero-, pre-vaccination: number analyzed (Participants) | 750 | 872
  HPV-16, sero-, pre-vaccination | 0 | 0
  HPV-16, sero-, Month 6: number analyzed (Participants) | 738 | 865
  HPV-16, sero-, Month 6 | 41 | 864
  HPV-16, sero-, Month 7: number analyzed (Participants) | 740 | 865
  HPV-16, sero-, Month 7 | 34 | 861
  HPV-16, sero-, Month 12: number analyzed (Participants) | 719 | 839
  HPV-16, sero-, Month 12 | 30 | 837
  HPV-16, sero-, Month 24: number analyzed (Participants) | 672 | 797
  HPV-16, sero-, Month 24 | 33 | 796
  HPV-16, sero-, Month 36: number analyzed (Participants) | 664 | 784
  HPV-16, sero-, Month 36 | 35 | 784
  HPV-16, sero-, Month 48: number analyzed (Participants) | 603 | 746
  HPV-16, sero-, Month 48 | 47 | 746
  HPV-16, sero+, pre-vaccination: number analyzed (Participants) | 147 | 164
  HPV-16, sero+, pre-vaccination | 147 | 164
  HPV-16, sero+, Month 6: number analyzed (Participants) | 139 | 162
  HPV-16, sero+, Month 6 | 119 | 161
  HPV-16, sero+, Month 7: number analyzed (Participants) | 139 | 163
  HPV-16, sero+, Month 7 | 106 | 162
  HPV-16, sero+, Month 12: number analyzed (Participants) | 134 | 154
  HPV-16, sero+, Month 12 | 101 | 154
  HPV-16, sero+, Month 24: number analyzed (Participants) | 138 | 146
  HPV-16, sero+, Month 24 | 96 | 146
  HPV-16, sero+, Month 36: number analyzed (Participants) | 127 | 142
  HPV-16, sero+, Month 36 | 88 | 142
  HPV-16, sero+, Month 48: number analyzed (Participants) | 118 | 145
  HPV-16, sero+, Month 48 | 85 | 145
  HPV-16, total, pre-vaccination: number analyzed (Participants) | 897 | 1036
  HPV-16, total, pre-vaccination | 147 | 164
  HPV-16, total, Month 6: number analyzed (Participants) | 877 | 1027
  HPV-16, total, Month 6 | 160 | 1025
  HPV-16, total, Month 7: number analyzed (Participants) | 879 | 1028
  HPV-16, total, Month 7 | 140 | 1023
  HPV-16, total, Month 12: number analyzed (Participants) | 853 | 993
  HPV-16, total, Month 12 | 131 | 991
  HPV-16, total, Month 24: number analyzed (Participants) | 810 | 943
  HPV-16, total, Month 24 | 129 | 942
  HPV-16, total, Month 36: number analyzed (Participants) | 791 | 926
  HPV-16, total, Month 36 | 123 | 926
  HPV-16, total, Month 48: number analyzed (Participants) | 721 | 891
  HPV-16, total, Month 48 | 132 | 891
  HPV-18, sero-, pre-vaccination: number analyzed (Participants) | 790 | 939
  HPV-18, sero-, pre-vaccination | 0 | 0
  HPV-18, sero-, Month 6: number analyzed (Participants) | 771 | 930
  HPV-18, sero-, Month 6 | 29 | 927
  HPV-18, sero-, Month 7: number analyzed (Participants) | 772 | 930
  HPV-18, sero-, Month 7 | 32 | 925
  HPV-18, sero-, Month 12: number analyzed (Participants) | 748 | 901
  HPV-18, sero-, Month 12 | 36 | 901
  HPV-18, sero-, Month 24: number analyzed (Participants) | 698 | 854
  HPV-18, sero-, Month 24 | 37 | 853
  HPV-18, sero-, Month 36: number analyzed (Participants) | 691 | 841
  HPV-18, sero-, Month 36 | 31 | 841
  HPV-18, sero-, Month 48: number analyzed (Participants) | 633 | 806
  HPV-18, sero-, Month 48 | 32 | 804
  HPV-18, sero+, pre-vaccination: number analyzed (Participants) | 108 | 97
  HPV-18, sero+, pre-vaccination | 108 | 97
  HPV-18, sero+, Month 6: number analyzed (Participants) | 105 | 97
  HPV-18, sero+, Month 6 | 90 | 96
  HPV-18, sero+, Month 7: number analyzed (Participants) | 105 | 97
  HPV-18, sero+, Month 7 | 90 | 97
  HPV-18, sero+, Month 12: number analyzed (Participants) | 106 | 92
  HPV-18, sero+, Month 12 | 89 | 92
  HPV-18, sero+, Month 24: number analyzed (Participants) | 102 | 89
  HPV-18, sero+, Month 24 | 84 | 89
  HPV-18, sero+, Month 36: number analyzed (Participants) | 98 | 86
  HPV-18, sero+, Month 36 | 73 | 86
  HPV-18, sero+, Month 48: number analyzed (Participants) | 91 | 86
  HPV-18, sero+, Month 48 | 70 | 86
  HPV-18, total, pre-vaccination | 108 | 97
  HPV-18, total, Month 6: number analyzed (Participants) | 876 | 1027
  HPV-18, total, Month 6 | 119 | 1023
  HPV-18, total, Month 7: number analyzed (Participants) | 877 | 1027
  HPV-18, total, Month 7 | 122 | 1022
  HPV-18, total, Month 12: number analyzed (Participants) | 854 | 993
  HPV-18, total, Month 12 | 125 | 993
  HPV-18, total, Month 24: number analyzed (Participants) | 800 | 943
  HPV-18, total, Month 24 | 121 | 942
  HPV-18, total, Month 36: number analyzed (Participants) | 789 | 927
  HPV-18, total, Month 36 | 104 | 927
  HPV-18, total, Month 48: number analyzed (Participants) | 724 | 892
  HPV-18, total, Month 48 | 102 | 890

22. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 ELISA Titers in the Immunogenicity Subset
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as ELISA Units per milliliter (EL.U/mL).
  GMTs are presented for the total group and also stratified according to initial (Month 0) HPV-16 or HPV-18 serostatus by ELISA [seronegative (sero-) or seropositive (sero+)].
Time Frame: At Months 6, 7, 12, 24, 36 and 48
Population: The analyses were performed on the ATP cohort for immunogenicity for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 898 | 1036
EL.U/mL
  Anti-HPV-16, sero-, pre-vaccination: number analyzed (Participants) | 750 | 872
  Anti-HPV-16, sero-, pre-vaccination | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  Anti-HPV-16, sero-, Month 6: number analyzed (Participants) | 738 | 865
  Anti-HPV-16, sero-, Month 6 | 4.4 [4.2 to 4.5] | 630.7 [591.6 to 672.4]
  Anti-HPV-16, sero-, Month 7: number analyzed (Participants) | 740 | 865
  Anti-HPV-16, sero-, Month 7 | 4.4 [4.2 to 4.6] | 9206.5 [8609.4 to 9845.1]
  Anti-HPV-16, sero-, Month 12: number analyzed (Participants) | 719 | 839
  Anti-HPV-16, sero-, Month 12 | 4.3 [4.2 to 4.4] | 3281.1 [3064.5 to 3513.0]
  Anti-HPV-16, sero-, Month 24: number analyzed (Participants) | 672 | 797
  Anti-HPV-16, sero-, Month 24 | 4.4 [4.2 to 4.5] | 1592.0 [1491.6 to 1699.2]
  Anti-HPV-16, sero-, Month 36: number analyzed (Participants) | 664 | 784
  Anti-HPV-16, sero-, Month 36 | 4.4 [4.2 to 4.5] | 1265.1 [1184.8 to 1350.8]
  Anti-HPV-16, sero-, Month 48: number analyzed (Participants) | 603 | 746
  Anti-HPV-16, sero-, Month 48 | 4.6 [4.4 to 4.8] | 1174.3 [1096.1 to 1258.0]
  Anti-HPV-16, sero+, pre-vaccination: number analyzed (Participants) | 147 | 164
  Anti-HPV-16, sero+, pre-vaccination | 29.7 [25.0 to 35.4] | 28.9 [24.7 to 33.8]
  Anti-HPV-16, sero+, Month 6: number analyzed (Participants) | 139 | 162
  Anti-HPV-16, sero+, Month 6 | 24.4 [19.9 to 29.8] | 1256.9 [1030.1 to 1533.7]
  Anti-HPV-16, sero+, Month 7: number analyzed (Participants) | 139 | 163
  Anti-HPV-16, sero+, Month 7 | 21.7 [17.4 to 27.0] | 6423.1 [5486.3 to 7520.0]
  Anti-HPV-16, sero+, Month 12: number analyzed (Participants) | 134 | 154
  Anti-HPV-16, sero+, Month 12 | 20.2 [16.3 to 25.1] | 2909.6 [2504.3 to 3380.4]
  Anti-HPV-16, sero+, Month 24: number analyzed (Participants) | 138 | 146
  Anti-HPV-16, sero+, Month 24 | 18.7 [15.0 to 23.2] | 1573.2 [1356.7 to 1824.2]
  Anti-HPV-16, sero+, Month 36: number analyzed (Participants) | 127 | 142
  Anti-HPV-16, sero+, Month 36 | 17.7 [14.0 to 22.2] | 1244.3 [1068.9 to 1448.4]
  Anti-HPV-16, sero+, Month 48: number analyzed (Participants) | 118 | 145
  Anti-HPV-16, sero+, Month 48 | 18.3 [14.5 to 23.0] | 1115.9 [959.6 to 1297.7]
  Anti-HPV-16, total, pre-vaccination: number analyzed (Participants) | 897 | 1036
  Anti-HPV-16, total, pre-vaccination | 5.6 [5.3 to 5.9] | 5.5 [5.2 to 5.8]
  Anti-HPV-16, total, Month 6: number analyzed (Participants) | 877 | 1027
  Anti-HPV-16, total, Month 6 | 5.7 [5.4 to 6.1] | 703.2 [659.5 to 749.7]
  Anti-HPV-16, total, Month 7: number analyzed (Participants) | 879 | 1028
  Anti-HPV-16, total, Month 7 | 5.6 [5.3 to 6.0] | 8695.7 [8171.9 to 9253.1]
  Anti-HPV-16, total, Month 12: number analyzed (Participants) | 853 | 993
  Anti-HPV-16, total, Month 12 | 5.5 [5.2 to 5.8] | 3220.5 [3026.4 to 3427.1]
  Anti-HPV-16, total, Month 24: number analyzed (Participants) | 810 | 943
  Anti-HPV-16, total, Month 24 | 5.6 [5.3 to 5.9] | 1589.1 [1497.2 to 1686.6]
  Anti-HPV-16, total, Month 36: number analyzed (Participants) | 791 | 926
  Anti-HPV-16, total, Month 36 | 5.4 [5.1 to 5.8] | 1261.9 [1188.3 to 1340.0]
  Anti-HPV-16, total, Month 48: number analyzed (Participants) | 721 | 891
  Anti-HPV-16, total, Month 48 | 5.7 [5.4 to 6.1] | 1164.6 [1093.9 to 1239.8]
  Anti-HPV-18, sero-, pre-vaccination: number analyzed (Participants) | 790 | 939
  Anti-HPV-18, sero-, pre-vaccination | 3.5 [3.5 to 3.5] | 3.5 [3.5 to 3.5]
  Anti-HPV-18, sero-, Month 6: number analyzed (Participants) | 771 | 930
  Anti-HPV-18, sero-, Month 6 | 3.7 [3.6 to 3.8] | 542.7 [510.2 to 577.2]
  Anti-HPV-18, sero-, Month 7: number analyzed (Participants) | 772 | 930
  Anti-HPV-18, sero-, Month 7 | 3.8 [3.6 to 3.9] | 4741.3 [4452.2 to 5049.1]
  Anti-HPV-18, sero-, Month 12: number analyzed (Participants) | 748 | 901
  Anti-HPV-18, sero-, Month 12 | 3.8 [3.7 to 3.9] | 1521.7 [1431.0 to 1618.1]
  Anti-HPV-18, sero-, Month 24: number analyzed (Participants) | 698 | 854
  Anti-HPV-18, sero-, Month 24 | 3.8 [3.7 to 3.9] | 704.4 [658.4 to 753.8]
  Anti-HPV-18, sero-, Month 36: number analyzed (Participants) | 691 | 841
  Anti-HPV-18, sero-, Month 36 | 3.7 [3.6 to 3.8] | 534.3 [498.9 to 572.1]
  Anti-HPV-18, sero-, Month 48: number analyzed (Participants) | 633 | 806
  Anti-HPV-18, sero-, Month 48 | 3.8 [3.7 to 3.9] | 476.2 [443.2 to 511.6]
  Anti-HPV-18, sero+, pre-vaccination: number analyzed (Participants) | 108 | 97
  Anti-HPV-18, sero+, pre-vaccination | 23.4 [18.9 to 29.1] | 24.8 [20.1 to 30.6]
  Anti-HPV-18, sero+, Month 6: number analyzed (Participants) | 105 | 97
  Anti-HPV-18, sero+, Month 6 | 19.6 [15.2 to 25.4] | 903.8 [714.0 to 1144.2]
  Anti-HPV-18, sero+, Month 7: number analyzed (Participants) | 105 | 97
  Anti-HPV-18, sero+, Month 7 | 20.8 [16.2 to 26.8] | 4135.7 [3548.6 to 4819.9]
  Anti-HPV-18, sero+, Month 12: number analyzed (Participants) | 106 | 92
  Anti-HPV-18, sero+, Month 12 | 19.9 [15.5 to 25.5] | 1509.5 [1271.3 to 1792.3]
  Anti-HPV-18, sero+, Month 24: number analyzed (Participants) | 102 | 89
  Anti-HPV-18, sero+, Month 24 | 18.9 [14.6 to 24.4] | 745.6 [620.1 to 896.6]
  Anti-HPV-18, sero+, Month 36: number analyzed (Participants) | 98 | 86
  Anti-HPV-18, sero+, Month 36 | 16.8 [12.8 to 22.1] | 580.9 [475.0 to 710.4]
  Anti-HPV-18, sero+, Month 48: number analyzed (Participants) | 91 | 86
  Anti-HPV-18, sero+, Month 48 | 16.5 [12.6 to 21.6] | 510.6 [415.7 to 627.2]
  Anti-HPV-18, total, pre-vaccination | 4.4 [4.2 to 4.6] | 4.2 [4.0 to 4.4]
  Anti-HPV-18, total, Month 6: number analyzed (Participants) | 876 | 1027
  Anti-HPV-18, total, Month 6 | 4.5 [4.3 to 4.8] | 569.5 [536.0 to 605.1]
  Anti-HPV-18, total, Month 7: number analyzed (Participants) | 877 | 1027
  Anti-HPV-18, total, Month 7 | 4.6 [4.4 to 4.9] | 4680.5 [4413.4 to 4963.7]
  Anti-HPV-18, total, Month 12: number analyzed (Participants) | 854 | 993
  Anti-HPV-18, total, Month 12 | 4.6 [4.4 to 4.9] | 1520.5 [1435.0 to 1611.2]
  Anti-HPV-18, total, Month 24: number analyzed (Participants) | 800 | 943
  Anti-HPV-18, total, Month 24 | 4.7 [4.4 to 4.9] | 708.2 [664.6 to 754.8]
  Anti-HPV-18, total, Month 36: number analyzed (Participants) | 789 | 927
  Anti-HPV-18, total, Month 36 | 4.5 [4.3 to 4.8] | 538.5 [504.7 to 574.5]
  Anti-HPV-18, total, Month 48: number analyzed (Participants) | 724 | 892
  Anti-HPV-18, total, Month 48 | 4.6 [4.3 to 4.8] | 479.4 [448.0 to 513.0]

23. Secondary Outcome: HPV-16 and HPV-18 Seroconversion (V5/J4 Monoclonal Inhibition Test)
Description: HPV-16 V5 cut-off was defined as greater than or equal to 41 ELU/mL. Only seronegative subjects were analysed. Seronegative subjects are subjects who had an antibody titer of less than 41 ELU/mL before vaccination.
  HPV-18 J4 cut-off was defined as greater than or equal to 110 EL.U/mL. Both seropositive and seronegative subjects were included in the analysis. Seropositive subjects were subjects with an antibody titer of greater than or equal to 110 EL.U/mL. Seronegative subjects were subjects with an antibody titer less than 110 EL.U/mL.
Time Frame: Month 0, 7, 12 and 24
Population: Analyses was performed on the Total Vaccinated Cohort on subjects with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 17 | 17
Participants
  pre-vaccination V5 HPV-16 | 0 | 0
  Month 7 V5 HPV-16 | 0 | 17
  Month 12 V5 HPV-16: number analyzed (Participants) | 5 | 2
  Month 12 V5 HPV-16 | 0 | 2
  Month 24 V5 HPV-16 | 0 | 17
  pre-vaccination J4 HPV-18 | 0 | 1
  Month 7 J4 HPV-18 | 0 | 17
  Month 12 J4 HPV-18: number analyzed (Participants) | 5 | 2
  Month 12 J4 HPV-18 | 1 | 1
  Month 24 V5 HPV-18 | 1 | 11

24. Secondary Outcome: HPV-16 and HPV-18 Geometric Mean Titers (GMT) (V5/J4 Monoclonal Inhibition Test)
Description: Titers were expressed as GMTs in ELISA units per milliliter (EL.U/mL).
Time Frame: Month 0, 7, 12, 24
Population: The analyses was performed on the Total Vaccinated cohort on subjects with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 17 | 17
EL.U/mL
  pre-vaccination V5 HPV-16 | 20.5 [20.5 to 20.5] | 20.5 [20.5 to 20.5]
  Month 7 V5 HPV-16 | 20.5 [20.5 to 20.5] | 816.7 [472.5 to 1411.4]
  Month 12 V5 HPV-16: number analyzed (Participants) | 5 | 2
  Month 12 V5 HPV-16 | 20.5 [20.5 to 20.5] | 173.5 [25.1 to 1199.3]
  Month 24 V5 HPV-16 | 20.5 [20.5 to 20.5] | 163.3 [104.0 to 256.6]
  pre-vaccination J4 HPV-18 | 55.0 [55.0 to 55.0] | 57.7 [52.1 to 63.8]
  Month 7 J4 HPV-18 | 55.0 [55.0 to 55.0] | 679.2 [423.6 to 1088.9]
  Month 12 J4 HPV-18: number analyzed (Participants) | 5 | 2
  Month 12 J4 HPV-18 | 71.0 [35.0 to 144.2] | 83.6 [0.4 to 17024.0]
  Month 24 V5 HPV-18 | 58.1 [51.7 to 65.2] | 139.5 [90.5 to 215.1]

25. Secondary Outcome: Number of Subjects Seropositive for Anti-HPV-16 and Anti-HPV-18 Antibodies Using Pseudovirion Based Neutralizing Assay (PBNA)
Description: Seropositivity was defined as subjects with a titer equal to or greater than 40.
  Subjects with an antibody titer smaller than 40 prior to vaccination were seronegative prior to vaccination and subjects with a titer equal to or greater than 40 were seropositive prior to vaccination.
Time Frame: At Month 0, 7, 12, 24, 36 and 48
Population: The analyses were performed on the ATP cohort for immunogenicity which included subjects for whom immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 47 | 48
Participants
  pre-vaccination HPV-16: number analyzed (Participants) | 44 | 46
  pre-vaccination HPV-16 | 0 | 0
  Month 7 HPV-16: number analyzed (Participants) | 44 | 46
  Month 7 HPV-16 | 0 | 46
  Month 12 HPV-16: number analyzed (Participants) | 43 | 45
  Month 12 HPV-16 | 0 | 45
  Month 24 HPV-16: number analyzed (Participants) | 40 | 46
  Month 24 HPV-16 | 0 | 46
  Month 36 HPV-16: number analyzed (Participants) | 33 | 41
  Month 36 HPV-16 | 0 | 41
  Month 48 HPV-16: number analyzed (Participants) | 33 | 41
  Month 48 HPV-16 | 0 | 40
  pre-vaccination HPV-18 | 0 | 0
  Month 7 HPV-18: number analyzed (Participants) | 44 | 46
  Month 7 HPV-18 | 0 | 46
  Month 12 HPV-18: number analyzed (Participants) | 43 | 45
  Month 12 HPV-18 | 0 | 44
  Month 24 HPV-18: number analyzed (Participants) | 40 | 46
  Month 24 HPV-18 | 0 | 46
  Month 36 HPV-18: number analyzed (Participants) | 33 | 41
  Month 36 HPV-18 | 0 | 41
  Month 48 HPV-18: number analyzed (Participants) | 33 | 41
  Month 48 HPV-18 | 2 | 39

26. Secondary Outcome: Titers for Anti-HPV-16 and Anti-HPV-18 Antibodies Using Pseudovirion Based Neutralizing Assay (PBNA)
Description: Titers were expressed as GMTs.
Time Frame: At month 0, 7, 12, 24, 36 and 48
Population: The analyses were performed on the ATP cohort for immunogenicity for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Havrix Group | Cervarix Group
Number analyzed (Participants) | 47 | 48
titer
  pre-vaccination HPV-16: number analyzed (Participants) | 44 | 46
  pre-vaccination HPV-16 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Month 7 HPV-16: number analyzed (Participants) | 44 | 46
  Month 7 HPV-16 | 20.0 [20.0 to 20.0] | 27364.8 [19780.1 to 37857.9]
  Month 12 HPV-16: number analyzed (Participants) | 43 | 45
  Month 12 HPV-16 | 20.0 [20.0 to 20.0] | 8385.9 [5857.3 to 12006.0]
  Month 24 HPV-16: number analyzed (Participants) | 40 | 46
  Month 24 HPV-16 | 20.0 [20.0 to 20.0] | 3647.4 [2586.5 to 5143.4]
  Month 36 HPV-16: number analyzed (Participants) | 33 | 41
  Month 36 HPV-16 | 20.0 [20.0 to 20.0] | 2245.1 [1616.6 to 3117.9]
  Month 48 HPV-16: number analyzed (Participants) | 33 | 41
  Month 48 HPV-16 | 20.0 [20.0 to 20.0] | 1931.1 [1294.4 to 2880.8]
  pre-vaccination HPV-18 | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Month 7 HPV-18: number analyzed (Participants) | 44 | 46
  Month 7 HPV-18 | 20.0 [20.0 to 20.0] | 9052.7 [6851.8 to 11960.5]
  Month 12 HPV-18: number analyzed (Participants) | 43 | 45
  Month 12 HPV-18 | 20.0 [20.0 to 20.0] | 1889.9 [1316.0 to 2714.1]
  Month 24 HPV-18: number analyzed (Participants) | 40 | 46
  Month 24 HPV-18 | 20.0 [20.0 to 20.0] | 1695.6 [1200.7 to 2394.4]
  Month 36 HPV-18: number analyzed (Participants) | 33 | 41
  Month 36 HPV-18 | 20.0 [20.0 to 20.0] | 1326.9 [948.0 to 1857.3]
  Month 48 HPV-18: number analyzed (Participants) | 33 | 41
  Month 48 HPV-18 | 23.8 [18.6 to 30.4] | 1078.1 [714.9 to 1625.6]

27. Secondary Outcome: Geometric Mean Titers of Anti-HPV-16 in Subjects Without and With 6-month Persistent Infection
Description: GMT for anti-HPV-16 antibodies by ELISA in subjects with breakthrough persistent infections 6-month definition, were compared to those in a matched set of subjects without breakthrough persistent infections. Due to the lack of seronegative subjects at Month 7, the hazard ratio (and Confidence Interval) was not calculated.
Time Frame: At Month 7
Population: The analysis was based on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available, only on subjects HPV-16 DNA negative and seronegative at baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Groups:
- Cervarix Group Without HPV-16 6-Month Persistent Infection: Subjects received 3 doses of Cervarix™ (GSK Biologicals' human papillomavirus [HPV] vaccine) at Months 0, 1 and 6 and who did not present 6-Month persistent infection with HPV-16.
- Cervarix Group With HPV-16 6-Month Persistent Infection: Subjects received 3 doses of Cervarix™ (GSK Biologicals' human papillomavirus [HPV] vaccine) at Months 0, 1 and 6, who presented 6-Month persistent infection with HPV-16.
Arm/Group | Cervarix Group Without HPV-16 6-Month Persistent Infection | Cervarix Group With HPV-16 6-Month Persistent Infection
Number analyzed (Participants) | 1123 | 45
EL.U/mL | 7667.34 [7212.13 to 8151.29] | 6986.30 [5692.83 to 8573.66]
Statistical Analysis 1: Comparison: Cervarix Group Without HPV-16 6-Month Persistent Infection vs Cervarix Group With HPV-16 6-Month Persistent Infection; Hazard ratio of anti-HPV-16 GMTs at Month 7 (by ELISA) in subjects without 6-month persistent infection compared to subjects with 6-month persistent infection; Test type: Superiority or Other; p = 0.3910, Chi-squared; Hazard Ratio (HR) = 0.798, 95% CI 2-sided [0.476 to 1.337]

28. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-16 Without and With 6-month Persistent Infection.
Description: Seroconversion rates for anti-HPV-16 antibodies by ELISA in subjects with breakthrough persistent infections 6-month definition, were compared to those in a matched set of subjects without breakthrough persistent infections. Due to the lack of seronegative subjects at Month 7, the hazard ratio (and Confidence interval) was not calculated.
Time Frame: At Month 7
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group Without HPV-16 6-Month Persistent Infection | Cervarix Group With HPV-16 6-Month Persistent Infection
Number analyzed (Participants) | 1123 | 45
Participants | 1118 | 45

29. Secondary Outcome: Geometric Mean Titers of Anti-HPV-16 in Subjects Without and With 12-month Persistent Infection
Description: GMTs for anti-HPV-16 antibodies by ELISA in subjects with breakthrough persistent infections 12-month definition, were compared to those in a matched set of subjects without breakthrough persistent infections.
Time Frame: At Month 7
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Groups:
- Cervarix Group Without HPV-16 12-Month Persistent Infection: Subjects received 3 doses of Cervarix™ (GSK Biologicals' human papillomavirus [HPV] vaccine) at Months 0, 1 and 6, without 12 Month persistent infection with HPV-16.
- Cervarix Group With HPV-16 12-Month Persistent Infection: Subjects received 3 doses of Cervarix™ (GSK Biologicals' human papillomavirus [HPV] vaccine) at Months 0, 1 and 6, with 12 Month persistent infection with HPV-16.
Arm/Group | Cervarix Group Without HPV-16 12-Month Persistent Infection | Cervarix Group With HPV-16 12-Month Persistent Infection
Number analyzed (Participants) | 1120 | 37
EL.U/mL | 7683.56 [7229.22 to 8166.44] | 6839.71 [5362.44 to 8723.96]
Statistical Analysis 1: Comparison: Cervarix Group Without HPV-16 12-Month Persistent Infection; Hazard ratio of anti-HPV-16 GMTs at Month 7 (by ELISA) in subjects without 12-month persistent infection compared to subjects with 12-month persistent infection; Test type: Superiority or Other; p = 0.3796, Chi-squared; Hazard Ratio (HR) = 0.778, 95% CI 2-sided [0.444 to 1.362]

30. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-16 Without and With 12-month Persistent Infection
Description: Seroconversion rates for anti-HPV-16 antibodies by ELISA in subjects with breakthrough persistent infections 12-month definition, were compared to those in a matched set of subjects without breakthrough persistent infections. Due to the lack of seronegative subjects at Month 7, the hazard ratio (and Confidence Interval) was not calculated.
Time Frame: At Month 7
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group Without HPV-16 12-Month Persistent Infection | Cervarix Group With HPV-16 12-Month Persistent Infection
Number analyzed (Participants) | 1120 | 37
Participants | 1115 | 37

31. Secondary Outcome: Geometric Mean Titers of Anti-HPV-18 in Subjects Without and With 6-month Persistent Infection
Description: GMTs for anti-HPV-18 antibodies by ELISA in subjects with breakthrough persistent infections 6-month definition, were compared to those in a matched set of subjects without breakthrough persistent infections.
Time Frame: At Month 7
Population: The analysis was based on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available, only on subjects HPV-18 DNA negative and seronegative at baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Groups:
- Cervarix Group Without HPV-18 6-Month Persistent Infection: Subjects received 3 doses of Cervarix™ (GSK Biologicals' human papillomavirus [HPV] vaccine) at Months 0, 1 and 6 and who did not present 6-Month persistent infection with HPV-18.
- Cervarix Group With HPV-18 6-Month Persistent Infection: Subjects received 3 doses of Cervarix™ (GSK Biologicals' human papillomavirus [HPV] vaccine) at Months 0, 1 and 6, who presented 6-Month persistent infection with HPV-18.
Arm/Group | Cervarix Group Without HPV-18 6-Month Persistent Infection | Cervarix Group With HPV-18 6-Month Persistent Infection
Number analyzed (Participants) | 1248 | 28
EL.U/mL | 3963.50 [3750.71 to 4188.37] | 2945.69 [2271.74 to 3819.58]
Statistical Analysis 1: Comparison: Cervarix Group Without HPV-18 6-Month Persistent Infection vs Cervarix Group With HPV-18 6-Month Persistent Infection; Hazard ratio of anti-HPV-18 GMTs at Month 7 (by ELISA) in subjects without 6-month persistent infection compared to subjects with 6-month persistent infection; Test type: Superiority or Other; p = 0.1035, Chi-squared; Hazard Ratio (HR) = 0.610, 95% CI [0.337 to 1.106]

32. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-18 Without and With 6-month Persistent Infection.
Description: Seroconversion rates for anti-HPV-18 antibodies by ELISA in subjects with breakthrough persistent infections 6-month definition, were compared to those in a matched set of subjects without breakthrough persistent infections. Due to the lack of seronegative subjects at Month 7, the hazard ratio (and Confidence Interval) was not calculated.
Time Frame: At Month 7
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group Without HPV-18 6-Month Persistent Infection | Cervarix Group With HPV-18 6-Month Persistent Infection
Number analyzed (Participants) | 1248 | 28
Participants | 1242 | 28

33. Secondary Outcome: Geometric Mean Titers of Anti-HPV-18 in Subjects Without and With 12-month Persistent Infection
Description: GMTs for anti-HPV-18 antibodies by ELISA in subjects with breakthrough persistent infections 12-month definition, were compared to those in a matched set of subjects without breakthrough persistent infections.
Time Frame: At Month 7
Population: as for outcome 31
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Groups:
- Cervarix Group Without HPV-18 12-Month Persistent Infection: Subjects received 3 doses of Cervarix™ (GSK Biologicals' human papillomavirus [HPV] vaccine) at Months 0, 1 and 6 and who did not present 12-Month persistent infection with HPV-18.
- Cervarix Group With HPV-18 12-Month Persistent Infection: Subjects received 3 doses of Cervarix™ (GSK Biologicals' human papillomavirus [HPV] vaccine) at Months 0, 1 and 6, who presented 12-Month persistent infection with HPV-18.
Arm/Group | Cervarix Group Without HPV-18 12-Month Persistent Infection | Cervarix Group With HPV-18 12-Month Persistent Infection
Number analyzed (Participants) | 1243 | 21
EL.U/mL | 3965.67 [3753.09 to 4190.29] | 3063.23 [2261.65 to 4148.91]
Statistical Analysis 1: Comparison: Cervarix Group Without HPV-18 12-Month Persistent Infection vs Cervarix Group With HPV-18 12-Month Persistent Infection; Hazard ratio of anti-HPV-18 GMTs at Month 7 (by ELISA) in subjects without 12-month persistent infection compared to subjects with 12-month persistent infection; Test type: Superiority or Other; p = 0.2111, Chi-squared; Hazard Ratio (HR) = 0.635, 95% CI 2-sided [0.312 to 1.293]

34. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-18 Without and With 12-month Persistent Infection
Description: Seroconversion rates for anti-HPV-18 antibodies by ELISA in subjects with breakthrough persistent infections 12-month definition, were compared to those in a matched set of subjects without breakthrough persistent infections. Due to the lack of seronegative subjects at Month 7, the hazard ratio (and Confidence Interval) was not calculated.
Time Frame: At Month 7
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group Without HPV-18 12-Month Persistent Infection | Cervarix Group With HPV-18 12-Month Persistent Infection
Number analyzed (Participants) | 1243 | 21
Participants | 1237 | 21

ADVERSE EVENTS:
Time Frame: Solicited symptoms during the 7-day post-vaccination period, Unsolicited AEs during the 30-day post-vaccination period, SAEs during the entire FU period.
Description: Results presented per group consist of a summary of the events (SAEs and AEs other than SAEs, respectively) reported, compiling overall number of subjects with events across the different periods of assessment.
Arm/Group | Havrix Group | Cervarix Group
Serious Adverse Events (participants affected / at risk) | 829/9325 | 835/9319
Other Adverse Events (participants affected / at risk) | 2678/9325 | 2869/9319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Havrix Group (N=9325) | Cervarix Group (N=9319)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 59 | 70
Appendicitis (Infections and infestations) | 59 | 46
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 40 | 54
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 46 | 43
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 27 | 20
Depression (Psychiatric disorders) | 19 | 20
Pyelonephritis (Infections and infestations) | 13 | 22
Premature labour (Pregnancy, puerperium and perinatal conditions) | 12 | 21
Abdominal pain (Gastrointestinal disorders) | 15 | 16
Pneumonia (Infections and infestations) | 10 | 20
Pyelonephritis acute (Infections and infestations) | 12 | 18
Gastroenteritis (Infections and infestations) | 14 | 14
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 8 | 18
Cholelithiasis (Hepatobiliary disorders) | 9 | 14
Ovarian cyst (Reproductive system and breast disorders) | 10 | 11
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 11 | 10
tonsillitis (Infections and infestations) | 8 | 13
Urinary tract infection (Infections and infestations) | 13 | 8
Suicide attempt (Psychiatric disorders) | 11 | 9
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 9 | 10
Road traffic accident (Injury, poisoning and procedural complications) | 10 | 9
Infectious mononucleosis (Infections and infestations) | 10 | 8
Pelvic inflammatory disease (Infections and infestations) | 5 | 13
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 7 | 9
Peritonsillar abscess (Infections and infestations) | 8 | 8
Ovarian cyst ruptured (Reproductive system and breast disorders) | 11 | 4
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 7 | 8
Acute tonsillitis (Infections and infestations) | 7 | 7
Concussion (Injury, poisoning and procedural complications) | 6 | 7
Gastritis (Gastrointestinal disorders) | 4 | 9
Ligament rupture (Injury, poisoning and procedural complications) | 10 | 3
Cholecystitis (Hepatobiliary disorders) | 4 | 6
Ankle fracture (Injury, poisoning and procedural complications) | 7 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Cellulitis (Infections and infestations) | 7 | 2
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 4 | 5
Joint dislocation (Injury, poisoning and procedural complications) | 7 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 5
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 3 | 6
Abdominal pain lower (Gastrointestinal disorders) | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3
Abortion induced (Surgical and medical procedures) | 3 | 5
Chronic tonsillitis (Infections and infestations) | 6 | 2
Endometriosis (Reproductive system and breast disorders) | 6 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 6 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 4
Foot fracture (Injury, poisoning and procedural complications) | 4 | 3
Head injury (Injury, poisoning and procedural complications) | 4 | 3
Hypersensitivity (Immune system disorders) | 5 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 3
Pregnancy induced hypertension (Pregnancy, puerperium and perinatal conditions) | 5 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1
Bipolar disorder (Psychiatric disorders) | 3 | 3
Cholecystitis acute (Hepatobiliary disorders) | 4 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 4
Dengue fever (Infections and infestations) | 3 | 3
Epilepsy (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 1 | 5
Major depression (Psychiatric disorders) | 5 | 1
Migraine (Nervous system disorders) | 2 | 4
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Overdose (Injury, poisoning and procedural complications) | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 2 | 3
Bronchitis (Infections and infestations) | 3 | 2
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 4
Deep vein thrombosis (Vascular disorders) | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Endometritis decidual (Infections and infestations) | 4 | 1
Premature baby (Pregnancy, puerperium and perinatal conditions) | 2 | 3
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 | 4
Psychotic disorder (Psychiatric disorders) | 3 | 2
Radius fracture (Injury, poisoning and procedural complications) | 3 | 2
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Bartholinitis (Reproductive system and breast disorders) | 2 | 2
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 1 | 3
Crohn's disease (Gastrointestinal disorders) | 3 | 1
Erysipelas (Infections and infestations) | 1 | 3
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 3
Limb injury (Injury, poisoning and procedural complications) | 2 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 3
Meningitis viral (Infections and infestations) | 1 | 3
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 2
Multiple sclerosis (Nervous system disorders) | 1 | 3
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Optic neuritis (Nervous system disorders) | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 3 | 1
Panic disorder (Psychiatric disorders) | 1 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 3 | 0
Anorexia nervosa (Psychiatric disorders) | 0 | 3
Appendicitis perforated (Infections and infestations) | 2 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 3
Colitis (Gastrointestinal disorders) | 2 | 1
Completed suicide (Psychiatric disorders) | 3 | 0
Convulsion (Nervous system disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Diverticulitis (Infections and infestations) | 1 | 2
Drug dependence (Psychiatric disorders) | 1 | 2
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 2
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Facial palsy (Nervous system disorders) | 1 | 2
Fallopian tube cyst (Reproductive system and breast disorders) | 0 | 3
Food allergy (Immune system disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Genital herpes (Infections and infestations) | 1 | 2
Hand fracture (Injury, poisoning and procedural complications) | 2 | 1
Homicide (Social circumstances) | 2 | 1
Infection (Infections and infestations) | 0 | 3
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Meningitis tuberculous (Infections and infestations) | 3 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 3 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 3
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Ovarian cyst torsion (Reproductive system and breast disorders) | 2 | 1
Peritonsillitis (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 1 | 2
Pilonidal cyst (Infections and infestations) | 2 | 1
Post abortion infection (Infections and infestations) | 2 | 1
Post procedural infection (Infections and infestations) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pyrexia (General disorders) | 1 | 2
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 1 | 2
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 2
Sinusitis (Infections and infestations) | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 3
Thermal burn (Injury, poisoning and procedural complications) | 2 | 1
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 3 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Tooth impacted (Gastrointestinal disorders) | 1 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Viral infection (Infections and infestations) | 2 | 1
Abortion induced incomplete (Injury, poisoning and procedural complications) | 2 | 0
Abortion infected (Infections and infestations) | 1 | 1
Accidental needle stick (Injury, poisoning and procedural complications) | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 1
Alcoholism (Psychiatric disorders) | 0 | 2
Anaphylactic shock (Immune system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 2
Bacterial infection (Infections and infestations) | 1 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 1
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Bronchopneumonia (Infections and infestations) | 2 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cervicitis (Infections and infestations) | 1 | 1
Chronic sinusitis (Infections and infestations) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Conversion disorder (Psychiatric disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Ear infection (Infections and infestations) | 2 | 0
Eating disorder (Psychiatric disorders) | 2 | 0
Endometritis (Infections and infestations) | 1 | 1
Epidemic nephropathy (Infections and infestations) | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 2 | 0
Gestational diabetes (Metabolism and nutrition disorders) | 1 | 1
Goitre (Endocrine disorders) | 1 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 2
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 2
Gynaecological chlamydia infection (Infections and infestations) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 2
Hepatitis a (Infections and infestations) | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 2
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 2
Kidney infection (Infections and infestations) | 0 | 2
Mastitis (Infections and infestations) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Parotitis (Infections and infestations) | 2 | 0
Parovarian cyst (Reproductive system and breast disorders) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia mycoplasmal (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 1
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Salmonellosis (Infections and infestations) | 1 | 1
Salpingitis (Infections and infestations) | 1 | 1
Salpingo-oophoritis (Infections and infestations) | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tooth abscess (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 1 | 1
Tubo-ovarian abscess (Infections and infestations) | 1 | 1
Typhoid fever (Infections and infestations) | 0 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Varicella (Infections and infestations) | 1 | 1
Vulvitis (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 0 | 2
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Abortion induced complete complicated (Injury, poisoning and procedural complications) | 0 | 1
Abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0
Acquired immunodeficiency syndrome (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Anoxic encephalopathy (Nervous system disorders) | 0 | 1
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Astrocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bacterial toxaemia (Infections and infestations) | 0 | 1
Bartholin's abscess (Infections and infestations) | 1 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 1
Benign intracranial hypertension (Nervous system disorders) | 1 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Bipolar ii disorder (Psychiatric disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 1 | 0
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone tuberculosis (Infections and infestations) | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0
Breast abscess (Infections and infestations) | 0 | 1
Breech extraction (Surgical and medical procedures) | 1 | 0
Bulimia nervosa (Psychiatric disorders) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0
Carcinoid tumour of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Cerebral toxoplasmosis (Infections and infestations) | 1 | 0
Chest pain (General disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1 | 0
Coeliac disease (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Colon injury (Injury, poisoning and procedural complications) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0
Device occlusion (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Diaphragmatic injury (Injury, poisoning and procedural complications) | 0 | 1
Dissociative disorder (Psychiatric disorders) | 0 | 1
Drowning (General disorders) | 0 | 1
Drug abuse (Psychiatric disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysthymic disorder (Psychiatric disorders) | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1
Emotional distress (Psychiatric disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1
Epiglottitis (Infections and infestations) | 1 | 0
Epstein-barr virus infection (Infections and infestations) | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Extrapulmonary tuberculosis (Infections and infestations) | 0 | 1
Eye infection toxoplasmal (Infections and infestations) | 0 | 1
Face presentation (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Faeces hard (Gastrointestinal disorders) | 1 | 0
False labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Fatigue (General disorders) | 0 | 1
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Foetal growth retardation (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Generalized anxiety disorder (Psychiatric disorders) | 1 | 0
Gestational trophoblastic tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glomerulonephritis acute (Renal and urinary disorders) | 0 | 1
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Haemorrhagic fever (Infections and infestations) | 1 | 0
Hepatitis c (Infections and infestations) | 0 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0
Herpes oesophagitis (Infections and infestations) | 1 | 0
Histrionic personality disorder (Psychiatric disorders) | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Hyperchromic anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Ileitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Induced abortion infection (Infections and infestations) | 1 | 0
Induced labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Infected bites (Infections and infestations) | 1 | 0
Infection parasitic (Infections and infestations) | 1 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intentional self-injury (Psychiatric disorders) | 1 | 0
Intestinal mass (Gastrointestinal disorders) | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ligament disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Malocclusion (Gastrointestinal disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 1
Meningitis pneumococcal (Infections and infestations) | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Migraine with aura (Nervous system disorders) | 1 | 0
Mouth cyst (Gastrointestinal disorders) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Nail operation (Surgical and medical procedures) | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephritis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Neuroborreliosis (Infections and infestations) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
obesity (Metabolism and nutrition disorders) | 0 | 1
Obstructed labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0
Ovarian abscess (Infections and infestations) | 0 | 1
Ovarian adhesion (Reproductive system and breast disorders) | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian torsion (Reproductive system and breast disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Panic reaction (Psychiatric disorders) | 1 | 0
Parotid abscess (Infections and infestations) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Peritoneal tuberculosis (Infections and infestations) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0
Placenta accreta (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Placenta praevia haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pleocytosis (Nervous system disorders) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Postpartum depression (Psychiatric disorders) | 0 | 1
Postpartum uterine subinvolution (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyoderma (Infections and infestations) | 1 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0
Renal colic (Skin and subcutaneous tissue disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Rhinitis hypertrophic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Snake bite (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Strabismus (Eye disorders) | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Sweat gland infection (Infections and infestations) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsillitis streptococcal (Infections and infestations) | 1 | 0
Tooth malformation (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 1
Trichomoniasis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 | 1
Uterine atony (Reproductive system and breast disorders) | 0 | 1
Uterine inversion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Uterine malposition (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Uterine perforation (Injury, poisoning and procedural complications) | 1 | 0
Uterine rupture (Injury, poisoning and procedural complications) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Vulval abscess (Infections and infestations) | 0 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Weight increased (Investigations) | 1 | 0
Whiplash injury (Injury, poisoning and procedural complications) | 1 | 0
Wolff-parkinson-white syndrome (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Havrix Group (N=9325) | Cervarix Group (N=9319)
Pain at injection site (General disorders) | 2403/3080 | 2787/3078
Redness at injection site (General disorders) | 851/3080 | 1349/3078
Swelling at injection site (General disorders) | 609/3080 | 1293/3078
Arthralgia (General disorders) | 551/3081 | 633/3078
Fatigue (General disorders) | 1652/3081 | 1771/3078
Fever ≥ 37.5 degrees Celsius (General disorders) | 342/3081 | 385/3078
Gastro-intestinal symptoms (General disorders) | 847/3081 | 856/3078
Headache (General disorders) | 1583/3081 | 1668/3078
Myalgia (General disorders) | 1381/3081 | 1607/3078
Rash (General disorders) | 258/3081 | 314/3078
Urticaria (General disorders) | 244/3081 | 300/3078
Headache (Nervous system disorders) | 250/3187 | 228/3184
Influenza (Infections and infestations) | 176/3187 | 157/3184
Gynaecological Chlamydia infection (Infections and infestations) | 1085 | 1035

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.